# PHASE 3, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED TRIAL TO EVALUATE EFFICACY AND SAFETY OF NITAZOXANIDE IN THE TREATMENT OF COLDS DUE TO ENTEROVIRUS/RHINOVIRUS INFECTION

PROTOCOL NO. RM08-3009

Study Sponsor:

The Romark Institute for Medical Research

Version: FINAL 2.0

December 23, 2020

#### STATEMENT OF COMPLIANCE

This study will be conducted in compliance with this protocol, current International Conference on Harmonization Good Clinical Practice (ICH GCP), United States (US) Code of Federal Regulations (CFR) applicable to clinical studies (45 CFR Part 46, 21 CFR 50, 21 CFR Part 312), and applicable regulatory requirements.

1

#### INVESTIGATOR'S AGREEMENT

#### CONFIDENTIALITY

The information in this protocol is provided to you, as an Investigator or consultant, for review by you, your staff, and an applicable institutional review committee. By accepting this document, you agree that information contained herein will be considered confidential and will not be disclosed to others, without written authority from The Romark Institute for Medical Research, except to the extent necessary to obtain: (a) Institutional Review Board approval and (b) informed consent from those persons to whom the investigational medicinal product will be administered.

#### APPROVAL OF FINAL PROTOCOL

My signature below constitutes agreement with this protocol. I am providing the necessary assurances that this study will be conducted by me and my staff according to all stipulations of the protocol, including all statements regarding confidentiality, and in complete accordance with all applicable regulations including current Good Clinical Practice guidelines and the ethical guidelines set by the World Medical Assembly (Declaration of Helsinki, last amendment in Fortaleza, Brazil October 2013). Furthermore, my signature below indicates that source documents will be available for review by the Sponsor or their designated representative.

| Principal Investigator Signature: | |
|--------------------------------------------------------|-----------|
| Principal Investigator | Date |
| Print name: | |
| With the signature below, the Sponsor approves of this | protocol. |
| Sponsor Signature: | |
| The Romark Institute for Medical Research | Date |
| Print name: | |

# TABLE OF CONTENTS

| STATE | MENT OF COMPLIANCE | 1 |
|--------|-------------------------------------------------------------|----|
| INVEST | ΓΙGATOR'S AGREEMENT | 2 |
| TABLE | OF CONTENTS | 3 |
| LIST O | F TABLES | 6 |
| LIST O | F FIGURES | 7 |
| 1. | PROTOCOL SUMMARY | 8 |
| 1.1. | Synopsis | 8 |
| 1.2. | Schedule of Assessments | 11 |
| 2. | INTRODUCTION | 12 |
| 2.1. | Enteroviruses/Rhinoviruses | 12 |
| 2.2. | Nitazoxanide (NTZ) | 13 |
| 2.2.1. | NTZ Inhibits Viral Replication and Cytokine Secretion | 13 |
| 2.2.2. | Pharmacokinetics of NTZ in Humans | 14 |
| 2.2.3. | Overview of Clinical Experience with NTZ | 15 |
| 2.2.4. | Early Clinical Experience with NTZ in Treatment of EV/RV | 16 |
| 2.2.5. | Study RM08-3005: NTZ in the Treatment of Colds Due to EV/RV | 16 |
| 2.3. | Rationale for the Study | 18 |
| 3. | STUDY OBJECTIVES | 18 |
| 4. | STUDY DESIGN | 18 |
| 4.1. | Study Design Overview | 18 |
| 4.2. | Rationale for Important Issues in the Study Design | 19 |
| 4.2.1. | Choice of NTZ Dose and Duration of Treatment | 19 |
| 4.2.2. | Choice of Control Group | 20 |
| 4.2.3. | Choice of Patient Population | 20 |
| 4.2.4. | Use of Vitamin B Complex Supplement | 21 |
| 4.2.5. | Choice of Patient-Reported Outcome Instrument | 22 |
| 4.2.6. | Choice of Primary Endpoint | 22 |
| 5. | STUDY POPULATION | 22 |
| 5.1. | Inclusion Criteria | 22 |
| 5.2. | Exclusion Criteria | 23 |
| 5.3. | Study Population Diversity | 24 |

| 6. | STUDY INTERVENTION | 24 |
|---|---|---|
| 6.1. | Study Intervention(s) Administration | 24 |
| 6.1.1. | Study Intervention Description | 24 |
| 6.1.2. | Dosing and Administration. | 25 |
| 6.2. | Preparation, Handling, Storage and Accountability | 25 |
| 6.2.1. | Acquisition and Accountability | 25 |
| 6.2.2. | Packaging and Labeling. | 25 |
| 6.3. | Randomization and Blinding | 26 |
| 6.4. | Study Intervention Compliance | 26 |
| 6.5. | Concomitant Therapy | 26 |
| 7. | STUDY INTERVENTION DISCONTINUATION AND PARTICIPANT DISCONTINUATION | 27 |
| 8. | STUDY PROCEDURES | 27 |
| 8.1. | Visit Procedures | 27 |
| 8.1.1. | Informed Consent | 27 |
| 8.1.2. | Medical History | 28 |
| 8.1.3. | Physical Examination | 28 |
| 8.1.4. | Body Measurements and Resting Vital Signs | 28 |
| 8.1.5. | Screening FLU-PRO | 29 |
| 8.1.6. | Randomization and Dispensing Study Medication. | 29 |
| 8.1.7. | Subject Instructions | 29 |
| 8.1.8. | Day 2-5 Subject Contact | 30 |
| 8.2. | Laboratory Assessments | 30 |
| 8.2.1. | Assessments in the Clinic | 30 |
| 8.2.2. | Central Laboratory Assessments | 31 |
| 8.2.3. | Pharmacokinetics Assessments | 31 |
| 8.2.4. | Plan for Monitoring Viral Resistance. | 31 |
| 8.3. | Subject Diary | 31 |
| 8.3.1. | Subject Diary Completion | 32 |
| 8.3.2. | Subject Diary Compliance Monitoring | 32 |
| 8.4. | Adverse Events and Serious Adverse Events | 32 |
| 8.4.1. | Definitions | 32 |
| 8.4.2. | Recording and Follow Up of Adverse Events | 33 |

| 8.4.3. | Reporting Requirement | 34 |
|---------------|--------------------------------------------------------|----|
| 8.4.4. | Medication Errors | 34 |
| 9. | STATISTICAL CONSIDERATIONS | 34 |
| 9.1. | Sample Size Determination | 34 |
| 9.2. | Efficacy Variables | 34 |
| 9.3. | Response Definitions | 35 |
| 9.3.1. | Response Definitions for the Primary Efficacy Analysis | 35 |
| 9.3.2. | Definitions for Complications of Colds | 36 |
| 9.4. | Statistical Methodology | 37 |
| 9.4.1. | Efficacy Analyses | 37 |
| 9.4.2. | Population Pharmacokinetics Analysis | 39 |
| 9.4.3. | Safety Analyses | 39 |
| 10. | OPERATIONAL CONSIDERATIONS | 39 |
| 10.1. | Regulatory, Ethical and Study Oversight Considerations | 39 |
| 10.1.1. | Ethics | 39 |
| 10.1.2. | Investigator Responsibilities | 40 |
| 10.1.3. | Quality Assurance and Quality Control | 40 |
| 10.1.4. | Safety Oversight | 40 |
| 10.1.5. | Data Handling and Record Keeping | 40 |
| 10.1.6. | Clinical Monitoring | 41 |
| 10.1.7. | Protocol Deviations | 41 |
| 10.1.8. | Study Discontinuation and Closure | 41 |
| 10.1.9. | Data and Report Requirements | 42 |
| 10.1.10. | Confidentiality and Privacy | 42 |
| 10.1.11. | Publication and Data Sharing | 42 |
| 10.1.12. | Key Roles and Study Governance | 42 |
| 11. | REFERENCES | 43 |
| APPEND | IX 1. PROTOCOL REVISION HISTORY | 46 |
| APPEND | IX 2. CONTACT INFORMATION | 50 |
| APPEND | IX 3. LIST OF ESSENTIAL DOCUMENTS FOR THE SITE | 51 |
| APPEND | IX 4. TOXICITY GRADING TABLES | 53 |
| <b>APPEND</b> | IX 5 FI II-PRO DOMAIN/SURDOMAIN STRUCTURE | 60 |

# LIST OF TABLES

| Table 1: | Schedule of Assessments | 11 |
|---|---|---|
| Table 2: | Summary of Tizoxanide and Tizoxanide Glucuronide Pharmacokinetics Parame | |
| Table 3: | Summary of Tizoxanide and Tizoxanide Glucuronide Trough Plasma Concentra (µg/mL) by Study Day | ations |
| Table 4: | Proportions of Subjects Experiencing Complications and Bronchitis for EV/RV Infected Subjects Enrolled in Study RM08-3005 | |
| Table 5: | Study Medication Label | 25 |
| Table 6: | Protocol Revision History | 46 |
| Table 7: | Study Contact Information | 50 |
| Table 8: | List of Essential Documents | 51 |
| Table 9: | Table for Clinical Abnormalities: Vital Signs | 53 |
| Table 10: | Table for Clinical Abnormalities: Systemic (General) | 54 |
| Table 11: | Table for Clinical Abnormalities: Systemic Illness | 54 |
| Table 12: | Table for Laboratory Abnormalities: Serum | 55 |
| Table 13: | Table for Laboratory Abnormalities: Hematology | 58 |
| Table 14: | Table for Laboratory Abnormalities: Urine | 59 |

# LIST OF FIGURES

| Figure 1: | Time to Sustained Response for EV/RV-Infected Subjects Enrolled in Study RM08- |
|---|---|
| | 3005 |

# 1. PROTOCOL SUMMARY

1.1. Synopsis

| 1.1. Synopsis | |
|---|---|
| Title of Study: | A Phase 3, Randomized, Double-Blind, Placebo Controlled Trial to Evaluate the Efficacy and Safety of Nitazoxanide in the Treatment of Colds Due to <i>Enterovirus/Rhinovirus</i> Infection |
| Name of Test Drug: Nitazoxanide 300 mg Tablets | |
| Name of Active Ingredient: | Nitazoxanide |
| Study Sponsor: | The Romark Institute for Medical Research |
| IND Number: | 140,445 |
| | STUDY DETAILS |
| Anticipated Study Period: | July 2020 – May 2021 |
| Protocol & Amendments: | Original Protocol: July 16, 2020<br>Version 2.0: December 23, 2020 |
| Investigators: | Multiple in the US |
| | OBJECTIVES |
| | nate the effect of NTZ in reducing the time to Sustained Response compared acebo in subjects with laboratory-confirmed EV/RV infection |
| secon | ate the proportion of subjects requiring systemic antibiotics for an infection ndary to EV/RV, including pneumonia, otitis media, bronchitis, sinusitis or yngitis |
| | Evaluate the proportion of subjects positive for EV/RV by PCR at each of Days 4 and 10 |
| i | Evaluate the proportion of subjects requiring systemic antibiotics for each infection secondary to EV/RV, including pneumonia, otitis media, bronchitis, sinusitis or pharyngitis |
| Safety Objective: Safet | ty will be assessed by analysis of adverse events. |
| | METHODOLOGY |
| Study Design: | Multicenter, randomized, double-blind trial |
| Treatments: | Subjects will be randomized 1:1 to one of the following groups: |
| | Group 1 (NTZ): Two NTZ 300 mg tablets b.i.d. for 5 days administered orally with food. |
| | Group 2 (Placebo): Two placebo tablets b.i.d. for 5 days administered orally with food. |
| Study Duration: | Subjects will receive 2 tablets b.i.d. for 5 days (10 doses). The follow up period will extend through the end of study visit at study Day 28. |
| | SUBJECT POPULATION |
| · | |

**Number of Subjects Planned:** At least 350 up to 400 subjects with laboratory-confirmed EV/RV infection. Data for subjects enrolled in concurrent study RM08-3008 (COVID-19 treatment study with the same selection criteria and procedures) with laboratory confirmed EV/RV infection at baseline will be allocated to this study for analysis and will count toward the 350 to 400 required subjects.

#### **Inclusion Criteria:**

- 1. Male or female at least 12 years of age
- 2. Presence of clinical signs and/or symptoms consistent with worsening or stable EV/RV infection (one of the following is required):
  - a. Presence of at least two respiratory symptom domains (head, throat, nose, chest, cough) with a score of ≥2 as determined by Screening FLU-PRO <u>OR</u>
  - b. Presence of at least one respiratory symptom domain (head, throat, nose, chest, cough) with a score of ≥2 as determined by Screening FLU-PRO with pulse rate ≥90 <u>OR</u>
  - c. Presence of at least one respiratory symptom domain (head, throat, nose, chest, cough) with a score of ≥2 as determined by Screening FLU-PRO with respiratory rate ≥16

<u>AND</u> patient reported assessment that symptoms are present, the symptoms are not consistent with the subject's usual health, the symptoms interfere with daily activities, and the symptoms have worsened or remained the same relative to the previous day, as confirmed by responses to questions in the Screening FLU-PRO.

- 3. Onset of symptoms no more than 72 hours before enrollment in the trial. Onset of symptoms is defined as the earlier of the first time at which the subject experienced subjective fever or any respiratory symptom (headache/head congestion, throat symptoms, nasal symptoms, chest symptoms, cough).
- 4. Willing and able to provide written informed consent (including assent by legal guardian if under 18 years of age) and comply with the requirements of the protocol, including completion of the subject diary and all protocol procedures.

#### **Exclusion Criteria:**

- 1. [Exclusion criterion removed in protocol version 2.0. See Revision History in Appendix1.]
- Subjects who experienced a previous episode of acute upper respiratory tract infection, otitis, bronchitis or sinusitis or received antibiotics for these conditions within two weeks prior to and including study day 1.
- 3. Severely immunodeficient persons including:
  - a. Subjects with immunologic disorders or receiving immunosuppressive therapy (e.g., for organ or bone marrow transplants, immunomodulatory therapies for certain autoimmune diseases)
  - b. Subjects with untreated HIV infection or treated HIV infection with a CD4 count below 350 cells/mm³ in the last six months
  - c. Subjects actively undergoing systemic chemotherapy or radiotherapy treatment for malignancy
  - d. Subjects using steroids as maintenance therapy for a chronic condition
- 4. Subjects with active respiratory allergies or subjects expected to require anti-allergy medications during the study period for respiratory allergies.
- 5. Females of childbearing potential who are either pregnant or sexually active without the use of birth control. Female subjects of child-bearing potential that are sexually active must have a negative baseline pregnancy test and must agree to continue an acceptable method of birth control for the duration of the study and for 1 month post-treatment. A double barrier method, oral birth control pills administered for at least 2 monthly cycles prior to study drug administration, an IUD, or medroxyprogesterone acetate

administered intramuscularly for a minimum of one month prior to study drug administration are acceptable methods of birth control for inclusion into the study. Female subjects are considered of childbearing potential unless they are postmenopausal (absence of menstrual bleeding for 1 year - or 6 months if laboratory confirmation of hormonal status), or have had a hysterectomy, bilateral tubular ligation or bilateral oophorectomy.

- 6. Subjects residing in the same household with another subject participating in the study.
- 7. Treatment with any investigational drug or vaccine therapy within 30 days prior to screening and willing to avoid them during the course of the study.
- 8. Receipt of any dose of NTZ within seven days prior to screening.
- 9. Known sensitivity to NTZ or any of the excipients comprising the study medication.
- 10. Subjects unable to swallow oral tablets or capsules.
- 11. Subjects with known severe heart, lung, neurological or other systemic disease that the Investigator believes could preclude safe participation.
- 12. Subjects likely or expected to require hospitalization unrelated to cold during the study period.
- 13. Subjects who, in the judgment of the Investigator, will be unlikely to comply with the requirements of this protocol including completion of the subject diary.
- 14. Subjects taking medications considered to be major CYP2C8 substrates. Refer to Table 6 in Section 6.5.
- 15. Persons with any clinical sign or symptoms suggestive of severe systemic illness with COVID-19, including the following:
  - a. shortness of breath at rest,
  - b. resting pulse ≥125 beats per minute,
  - c. resting respiratory rate  $\geq 30$  breaths per minute, or
  - d.  $SpO_2 \le 93\%$  on room air at sea level.
- 16. Subjects known to have a diagnostic test positive for SARS-CoV-2 or influenza infection within the preceding three weeks.

#### **ASSESSMENTS**

#### Efficacy:

- Subjects will complete a diary recording oral temperature twice daily and the FLU-PRO® patient reported outcomes instrument once daily in the evening for 21 days for efficacy evaluation.
- Subjects will be contacted daily by site staff on study days 2-7 to screen for progression to severe
  illness or other complications.

**Virology:** Nasopharyngeal swab samples will be collected on each of study Days 1, 4 and 10 for analysis of virology endpoints.

**Safety:** The safety of study drug administration will be monitored by assessment of adverse events from baseline through the Day 28 study exit, clinical laboratory testing at baseline and on Day 10, physical examinations and vital signs assessments at screening, Day 10 and Day 22 and telephone monitoring/at home visits during Day 2 through Day 7 and Day 28.

**Pharmacokinetics:** On the morning of Day 4 prior to dosing, trough plasma samples will be collected.

# 1.2. Schedule of Assessments

**Table 1:** Schedule of Assessments

| | Screening | Baseline | Treatment Period | Diary Period | Follow-Up Visits | | | Unscheduled | |
|---|---|---|---|---|---|---|---|---|---|
| Assessment | Day 1 | Day 1 | Day 2-7 | Day 1-21 | Day<br>4±1 | Day<br>10±3 | Day 22+3 | Day 28+3 | As Needed |
| Signed informed consent/assent <sup>1</sup> | X | | | | | | | | |
| Demographics, smoking & medical history <sup>2</sup> | X | | | | | | | | |
| Urine pregnancy test <sup>7</sup> | X | | | | | | | | |
| Physical examination <sup>3</sup> | X | | | | X <sup>4</sup> | X <sup>4</sup> | $X^4$ | | $X^4$ |
| Body weight and resting vital signs <sup>5</sup> | X | | | | X | X | X | | X |
| Complete Screening FLU-PRO <sup>6</sup> | X | | | | | | | | |
| Evaluate eligibility <sup>7</sup> | X | | | | | | | | |
| Collect nasopharyngeal swabs <sup>8</sup> | | X | | | X | X | | | |
| Collect blood sample for lab safety tests <sup>8</sup> | | X | | | | | X | | X |
| Collect blood sample for antibody tests <sup>8</sup> | | X | | | | | X | | |
| Collect blood sample for pharmacokinetics <sup>8</sup> | | | | | X | | | | |
| Collect urine sample for routine urinalysis <sup>8</sup> | | X | | | | | X | | X |
| Record concomitant medications | | X | | | X | X | X | | X |
| Randomize & dispense study medication <sup>9</sup> | | X | | | | | | | |
| First dose and practice diary in-office <sup>9,10</sup> | | X | | | | | | | |
| Review/record adverse events <sup>11</sup> | | X | | | X | X | X | | X |
| Instructions re: dosing, concomitant medications, diary completion, follow-up visits, and emergency care <sup>12</sup> | | X | X | | X | X | X | | X |
| Contact subject to screen for complications | | | X <sup>13</sup> | | | | | X <sup>14</sup> | |
| Complete diary (subject responsibility) <sup>10</sup> | | | | X | | | | | |
| Review subject diary entries (site responsibility) <sup>15</sup> | | | and Continue 1 | X | | | Can Continu 9 | | Pag Section 5.0 |

<sup>&</sup>lt;sup>1</sup> See Section 8.1.1

<sup>&</sup>lt;sup>2</sup> See Section 8.1.2

<sup>&</sup>lt;sup>3</sup> See Section 8.1.3

<sup>&</sup>lt;sup>4</sup> Completed as necessary, see Section 8.1.3

<sup>&</sup>lt;sup>5</sup> See Section 8.1.4

<sup>&</sup>lt;sup>6</sup> See Section 8.1.5

<sup>&</sup>lt;sup>7</sup> See Section 5.0

<sup>&</sup>lt;sup>8</sup> See Section 8.2

<sup>&</sup>lt;sup>11</sup> See Section 8.4

<sup>&</sup>lt;sup>12</sup> See Section 8.1.7

<sup>&</sup>lt;sup>13</sup> See Section 8.1.8

<sup>&</sup>lt;sup>14</sup> See Section 8.1.9

#### 2. INTRODUCTION

#### 2.1. Enteroviruses/Rhinoviruses

There are more than 500 million non-influenza viral respiratory infections or "common colds" each year in the United States, with adults experiencing as many as 2-6 illnesses per year and children experiencing 6-8 (Fendrick et al. 2003, Turner 1997, Worrall 2011).

Colds have been reported to account for as much as 40% of time lost from work in the employed population and 30% of school absences (Kirkpatrick 1996). In a study conducted from November of 2000 to February of 2001, the total economic impact of non-influenza viral respiratory tract infections was nearly \$40 billion (Fendrick et al. 2003). Adjusted for inflation (February 2001 to January 2018), the economic impact today would exceed \$56 billion (USDOL Bureau of Labor Statistics 2018).

Fifty (50) to 67% of non-influenza viral respiratory tract infections are associated with viruses from the genus Enterovirus (EV), which belong to the Picornaviridae family (Atkinson et al. 2016). Within the EV genus, there are presently fifteen species including Rhinovirus A, Rhinovirus B, Rhinovirus C and Enterovirus A through L (The Pirbright Institute 2018). There are hundreds of EV serotypes, preventing the development of an effective vaccine or production of sufficient individual immunity to avoid multiple infections annually (Jacobs et al. 2013). A large majority of respiratory tract infections caused by viruses from the Enterovirus genus are due to Rhinovirus species, and RT-PCR assays do not distinguish between the different species of enteroviruses. Therefore, in this document we will refer to these viruses as Enterovirus/Rhinovirus (EV/RV).

EV/RV infection has been described as a "cytokine disease" because infection is characterized by massive upregulation of IFN, IL-1, IL-6, IL-8, TNF-α, granulocyte macrophage colony-stimulating factor and RANTES (Atkinson et al. 2016). Common symptoms include rhinorrhea, nasal congestion, sore throat, cough, headache, fever, and malaise. A natural history study of EV/RV infections demonstrated that patients were able to self-diagnose a cold in less than a day, with most patients self-diagnosing less than 8 hours from symptom onset (Arruda et al. 1997).

Colds due to EV/RV infection are generally considered self-limiting and do not cause respiratory distress. With advances in viral detection methods, however, colds due to EV/RV infection have been linked to exacerbations of COPD, asthma development, severe bronchiolitis in pediatric patients, and fatal pneumonia in elderly and immunocompromised adults. These severe outcomes are in addition to the milder commonly accepted complications of the common cold including secondary otitis media, sinusitis, pneumonia, and, in pediatric patients, croup and bronchiolitis (Jacobs et al. 2013).

Because there are no FDA-approved antiviral drugs for treatment of colds due to EVs, the standard of care is treatment of symptoms with over-the-counter (OTC) symptom relief medication including antihistamines, decongestants, analgesics, antitussives, NSAIDs, and combinations thereof. Most of these treatments have not shown clear benefit (Allan and Arroll 2014). Antiviral drugs to mitigate the impact of EV/RV infection are therefore needed.

# 2.2. Nitazoxanide (NTZ)

NTZ is a thiazolide anti-infective with *in vitro* activity against parasites, anaerobic bacteria, and viruses (Anderson and Curran 2007).

ALINIA® (NTZ) for Oral Suspension (patients 1 year of age and older) and ALINIA (NTZ) Tablets (patients 12 years and older) are marketed in the United States for the treatment of diarrhea caused by *Giardia lamblia* or *Cryptosporidium parvum*. ALINIA for Oral Suspension and ALINIA Tablets have not been shown to be superior to placebo for the treatment of diarrhea caused by *Cryptosporidium parvum* in HIV-infected or immunodeficient patients (ALINIA Prescribing Information 2019).

# 2.2.1. NTZ Inhibits Viral Replication and Cytokine Secretion

Tizoxanide, the active circulating metabolite of NTZ, has been shown to possess antiviral activity in cell culture against a broad range of viruses including influenza A and B viruses, coronaviruses (SARS-CoV-2, MERS-CoV, HCoV-229E, HCoV-OC43, HCoV-NL63, canine CoV S-378, murine coronavirus, mouse hepatitis virus strain A59 (MHV-A59)), parainfluenza (Sendai) virus, RSV A-2, rotavirus, norovirus, hepatitis C virus genotypes 1a and 1b, Japanese encephalitis virus, dengue fever virus-2, yellow fever virus, hepatitis B virus, and human immunodeficiency virus (HIV) (Rossignol 2014, Rossignol 2016, Wang et al. 2020, Piacentini et al. 2018, Romark data on file). Experiments in HeLa R19 cells have shown that NTZ inhibits replication of rhinovirus A serotypes 2 and 16 (Romark Study Report RM01-0434). Concentrations of tizoxanide required to inhibit replication of these viruses by 50% (EC50s) were generally between 0.2 and 3  $\mu$ M depending upon the test conditions.

The anti-influenza activity of nitazoxanide and its circulating metabolite, tizoxanide, has been investigated in human (Monocytic U937, T-lymphocytic Jurkat, and Alveolar type II-like A549) and canine (MDCK) cells after infection with multiple different strains of influenza A virus including oseltamivir-resistant and amantadine-resistant strains (Rossignol et al. 2009, Ashton et al. 2010, Sleeman et al. 2014). In a study of the susceptibility of 210 circulating seasonal influenza viruses to tizoxanide demonstrated median EC50 values ( $\pm$ IQR) of 0.48  $\mu$ M (0.33-0.71), 0.62  $\mu$ M (0.56-0.75), 0.66  $\mu$ M (0.62-0.69), and 0.60  $\mu$ M (0.51-0.67) for A (H1N1)pdm09, A (H3N2), B (Victoria lineage) and B (Yamagata lineage), respectively (Tilmanis et al. 2017).

Laboratory studies to evaluate the potential for resistance of influenza A virus to tizoxanide have been unable to select for resistant virus (Romark Study Report RM01-0417). These studies suggest a low potential for resistance.

Studies in peripheral blood mononuclear cells have also shown tizoxanide suppresses secretion of pro-inflammatory cytokines that are upregulated by viral respiratory infections (VRIs). Concentrations required to suppress cytokine secretion by 50% for IL-2, IL-4, IL-5, IL-6, IL-8, IL-10 and TNF- $\alpha$  ranged from 2.0 to 9.8  $\mu$ M (Rossignol and van Baalen 2018, Romark Study Report 9264). Nitazoxanide has also been shown to suppress IL-6 production in thioglycollate broth-injected mice (Hong et al. 2012).

Ongoing studies of the mechanism of action of NTZ have shown NTZ and tizoxanide modulate mitochondrial function by uncoupling oxidative phosphorylation. Studies indicate tizoxanide decreases cellular ATP in a dose-dependent manner in MDCK cells and in MDCK cells infected with influenza viruses. Maximum inhibition of ATP in influenza-infected or uninfected MDCK

cells reaches up to 45% after 24 hours of exposure to 100  $\mu$ M tizoxanide. In these experiments, a 10% reduction of ATP achieved by adding less than 10  $\mu$ M tizoxanide is sufficient to inhibit influenza virus replication by approximately 90%. The decrease in cellular ATP does not affect cell viability and is reversible after eliminating tizoxanide from the culture (Rossignol and van Baalen 2018). Studies of a number of different viruses have shown viral replication is ATP-dependent (Braakman et al. 1992, Braakman et al. 1991, Doms et al. 1987, Chang et al. 2009, Mirazimi and Svensson 2000). In the case of NTZ, key viral proteins like hemagglutinin (influenza), F-protein (RSV and parainfluenza), and N protein (coronavirus) have been identified as potential end targets of this mechanism (Rossignol et al. 2009, Piacentini et al. 2018, Cao et al. 2015). In addition, inhibition of ATP and its downstream effect on AMP-activated protein kinase activation has been shown to suppress secretion of pro-inflammatory cytokines (Lee et al. 2017, Sag et al. 2008, Wang et al. 2003).

The activity of NTZ in inhibiting replication of a broad range of respiratory viruses as well as the secretion of pro-inflammatory cytokines upregulated during respiratory virus infection has prompted clinical development of NTZ for treatment or prophylaxis of respiratory illness caused by VRIs.

#### 2.2.2. Pharmacokinetics of NTZ in Humans

NTZ is not detectable in the plasma following oral administration of the drug. The main metabolites of NTZ in humans are tizoxanide and tizoxanide glucuronide. Tizoxanide is highly bound to plasma proteins (>99%). The absorption of NTZ in immediate release tablets is significantly enhanced (Cmax and AUC of tizoxanide and tizoxanide glucuronide in plasma are more than doubled) when it is administered with food. In fasted human volunteers receiving a single 500 mg dose of 14C NTZ, approximately one-third of the dose was excreted in urine as tizoxanide and tizoxanide glucuronide, and two-thirds was excreted in feces as tizoxanide. No other significant metabolites were detected (NT-300 COVID/VRI-Investigators Brochure).

The pharmacokinetics of tizoxanide and tizoxanide glucuronide during repeated oral dosing of NTZ 300 mg extended release tablets administered 600 mg twice daily with food were evaluated in healthy volunteers. Twelve (12) subjects received two NTZ controlled release tablets twice daily with food for 7 days. The pharmacokinetics were studied in plasma up to 12 hours post-dose after the morning dose on Day 1 and Day 7, and before the morning dose on Day 2-6. Based on mixed effect analysis of variance, the steady state tizoxanide and tizoxanide glucuronide plasma concentrations was reached by Day 2, after one day of treatment with NTZ at 600 mg b.i.d. The main pharmacokinetics parameters of tizoxanide and tizoxanide glucuronide are summarized in the table below:

Table 2: Summary of Tizoxanide and Tizoxanide Glucuronide Pharmacokinetics
Parameters

| PK Parameter (unit) | Tizox | anide | Tizoxanide Glucuronide | |
|---|---|---|---|---|
| | Day 1 | Day 7 | Day 1 | Day 7 |
| | N=12 | N=12 | N=12 | N=12 |
| Cmax (µg/mL) | $5.23 \pm 2.71$ | $8.16 \pm 4.16$ | $4.88 \pm 1.72$ | $8.96 \pm 3.48$ |
| tmax (h) | 6.00 (4.00-9.00) | 5.00 (3.00-8.00) | 6.00 (5.00-11.00) | 5.50 (0.00-7.02) |

| PK Parameter (unit) | Tizox | anide | Tizoxanide Glucuronide | |
|---|---|---|---|---|
| tlag (h) | 0.00 (0.00-2.00) | 0.00 (0.00-0.00) | 0.50 (0.00-2.00) | 0.00 (0.00-0.00) |
| AUC0-t (μg.h/mL) | $26.9 \pm 16.1$ | $52.5 \pm 33.7$ | $29.5 \pm 12.1$ | $75.0 \pm 37.8$ |
| AUC0- T (μg.h/mL) | $28.6 \pm 16.3^{a}$ | $48.3\pm31.9^b$ | $30.5 \pm 12.2^{\circ}$ | $75.2 \pm 37.9$ |
| C T (µg/mL) | $0.709 \pm 0.987$ | $1.72 \pm 2.04$ | $1.39 \pm 0.846$ | $3.89 \pm 2.88$ |
| AUC0-∞ (μg.h/mL) | $27.8 \pm 17.8^{b}$ | $52.3 \pm 35.6^{b}$ | $35.3\pm16.5^{\text{d}}$ | $62.1 \pm 24.2^{e}$ |
| t1/2 (h) | $1.66 \pm 0.408^{b}$ | $2.19 \pm 0.485^{b}$ | $2.70 \pm 0.848^{c}$ | $4.99 \pm 5.20$ |
| λz (1/h) | $0.441 \pm 0.106^{b}$ | $0.331 \pm 0.0733^{b}$ | $0.282 \pm 0.0902^{c}$ | $0.201 \pm 0.0813$ |
| Cavg (µg/mL) | NA | $4.02 \pm 2.66$ b | NA | $6.27 \pm 3.16$ |
| Cmin (µg/mL) | NA | $1.50 \pm 1.83$ | NA | $3.63 \pm 3.00$ |
| PTF (%) | NA | $193 \pm 39.1b$ | NA | $101 \pm 40.7$ |
| Swing (%) | NA | $1039 \pm 656$ | NA | $268 \pm 194$ |

Values are arithmetic mean  $\pm$  SD, except median (range) for  $t_{max}$  and  $t_{lag}$ 

Table 3: Summary of Tizoxanide and Tizoxanide Glucuronide Trough Plasma Concentrations (μg/mL) by Study Day

| Analyte | Day 1 | Day 2 | Day 3 | Day 4 | Day 5 | Day 6 | Day 7 |
|-------------|-------|-------|-------|-------|-------|-------|-------|
| Tizoxanide | 0.709 | 1.55 | 2.36 | 3.24 | 3.80 | 3.26 | 3.02 |
| | (139) | (100) | (101) | (100) | (146) | (119) | (99) |
| Tizoxanide | 1.39 | 3.68 | 4.38 | 5.35 | 5.83 | 5.94 | 5.65 |
| Glucuronide | (61) | (72) | (73) | (77) | (99) | (91) | (69) |

#### 2.2.3. Overview of Clinical Experience with NTZ

NTZ has been marketed for diarrheal disease caused by *Giardia* or *Cryptosporidium* in the United States since 2003 and in Latin America since 1996. It is estimated that more than 350 million patients have been exposed to NTZ worldwide. No drug-related serious adverse events have been reported during post-marketing experience with NTZ.

Over 7,500 subjects have been treated with NTZ in clinical trials, including 3,147 subjects 12 years of age and older who have been exposed to the NTZ 300 mg extended release tablets (as monotherapy, n = 2,659, or in combination with oseltamivir, n = 488). Of the 3,147 subjects, 2,659 were given a dose of 600 mg twice daily for 5 days. The most commonly (at least 2% of treated subjects) reported adverse events (AEs) regardless of causality assessment were: chromaturia (10.8%), diarrhea (6.3%), abdominal pain/abdominal pain upper/abdominal pain lower (2.8%), bronchitis (2.8%), nausea (2.7%), and headache (2.3%). In the placebo-controlled trials, the rates of occurrence of AEs did not differ significantly from those of placebo except for

N = number of subjects with data; NA = not applicable

<sup>&</sup>lt;sup>a</sup> N=10; <sup>b</sup> N=11; <sup>c</sup> N=11; <sup>d</sup> N=8; <sup>e</sup> N=7

chromaturia (10.8% compared to 0.8% for placebo). Less than 1% of subjects discontinued therapy because of AEs (NT-300 Investigators Brochure-COVID/VRI).

#### 2.2.4. Early Clinical Experience with NTZ in Treatment of EV/RV

Subjects with laboratory-confirmed EV/RV infection were enrolled in two phase 3 randomized placebo-controlled clinical trials of NTZ for the treatment of influenza. Subjects presented to the clinic with oral temperatures ≥100.4°F and at least one respiratory and one constitutional symptom. Subjects assessed seven symptoms as absent, mild, moderate or severe twice daily for at least seven days (study RM08-3001) or at least 14 days (study RM08-3002) and up to 28 days. The primary endpoint for both studies was Time to Alleviation of Symptoms, defined as all symptoms rated absent or mild for at least 21.5 hours, for subjects with laboratory-confirmed influenza infection. This analysis was repeated for subjects with laboratory-confirmed EV/RV infection as exploratory analyses.

Study RM08-3001 was a dose-ranging study comparing NTZ 600 mg and NTZ 300 mg to placebo. Eighty-eight (88) subjects with EV/RV as the sole identified pathogen were enrolled (n=29, 33 and 26 in the NTZ 600 mg, NTZ 300 mg, and placebo groups, respectively). No differences in times to alleviation of symptoms were observed across treatment groups [Median (IQR): 105.1 (60-159) for the 600 mg NTZ group, 86.7 (70-119) for the 300 mg NTZ group, and 90.8 (59-134) for the placebo group].

Study RM08-3002 was a factorial trial of NTZ 600 mg and oseltamivir (OST). The study enrolled 228 subjects with EV/RV as the sole infection at baseline (n=55, 51, 61 and 61 for the NTZ, OST, NTZ+OST and placebo groups, respectively). Subjects treated with NTZ monotherapy had 31-hour treatment benefit at the median compared to placebo treated subjects [Median (IQR): 115.6 (69-210) for the NTZ group, 146.5 (92-298) for the placebo group, p=0.0390 for the Wilcoxon test and p=0.0128 for the Log Rank test).

The seven-symptom scale used in studies RM08-3001 and RM08-3002, though used in nearly every historical study of outpatient antivirals for viral respiratory infection, has not demonstrated content validity nor context validity and lacks internal consistency reliability, leading to inconsistent results across clinical trials, including studies of approved antivirals such as oseltamivir. The results of studies RM08-3001 and RM08-3002 formed the hypothesis that was the basis of study RM08-3005: that treatment benefit could be demonstrated for NTZ compared to placebo in subjects with laboratory-confirmed EV/RV infection with the use of an appropriately developed and validated patient reported outcomes (PRO) instrument and meaningful analysis methodology.

#### 2.2.5. Study RM08-3005: NTZ in the Treatment of Colds Due to EV/RV

Study RM08-3005 was a randomized placebo-controlled study of NTZ in the treatment of colds due to EV/RV. Subjects completed a daily diary for 21 days including the FLU-PRO instrument, a symptoms questionnaire with established content validity, context validity, reliability and responsiveness to change. Five-hundred eighty-four (584) subjects with laboratory-confirmed EV/RV infection were enrolled. The methodology for deriving the symptom response definition was intended to correlate symptom ratings to subject assessments of usual health status (a yes/no global assessment question in FLU-PRO). Median (IQR) Times to Return to Usual Health were 154.1 (80-320) and 174.9 (104-345) hours for the NTZ and placebo groups, respectively

(p=0.0712). While the time of symptom response and time of return to usual health were moderately correlated (r=0.43), the methodology returned a time of symptom response that was, on average, 4.5 study days from the time of return to usual health as reported by the subject, indicating that the methodology used to derive the symptom response definition should be optimized.

An improved symptom response definition (Sustained Response, see Section 9.3) was developed based on this data and is proposed for use in the present study. Applying this response definition and the patient selection criteria proposed for the present study, NTZ-treated subjects with laboratory-confirmed EV/RV infection experienced a treatment benefit of 101 hours at the median in Time to Sustained Response [Median (IQR): 151.0 (81-367) for the NTZ group, 252.0 (126->504) for the placebo group, p=0.0002 for the Wilcoxon test and p=0.0004 for the Log Rank test]. See Figure 1 below for Kaplan-Meier curves of Time to Sustained Response for this population.

Figure 1: Time to Sustained Response for EV/RV-Infected Subjects Enrolled in Study RM08-3005



The proportion of NTZ-treated EV/RV-infected subjects experiencing any complication was 40% lower than the proportion of EV/RV-infected subjects experiencing any complication in the placebo group. The proportion of NTZ-treated EV/RV-infected subjects experiencing bronchitis (the most frequent complication observed in this population) was 67% lower than for EV/RV-infected subjects randomized to the placebo group (see Table 4 below).

Table 4: Proportions of Subjects Experiencing Complications and Bronchitis for EV/RV-Infected Subjects Enrolled in Study RM08-3005

| Complication | NTZ<br>(N=286) | Placebo<br>(N=298) | <i>P</i> -value |
|---|---|---|---|
| Subjects experiencing any complication of EV/RV infection | 12 (4%) | 20 (7%) | 0.2057 |
| Subjects diagnosed with bronchitis | 3 (1%) | 9 (3%) | 0.1429 |

Subjects treated with NTZ were also significantly less likely to have EV/RV detected by RT-PCR in nasopharyngeal swabs collected on study day 7 (188/283, 66% vs 223/294, 76%, p=0.0132)

Treatment with 600 mg NTZ b.i.d. for five days was well tolerated by all subjects. The most frequently reported TEAEs (≥2% in any treatment group) were chromaturia (n=153 in the NTZ group and n=10 in the placebo group, p<0.0001,), diarrhoea (n=53 in the NTZ group, n=38 in the placebo group, NS), and nausea (n=24 in the NTZ group, n=19 in the placebo group, NS). Frequency and severity of adverse events were similar across treatment groups except for chromaturia, which was mild and more frequent in the NTZ group.

# 2.3. Rationale for the Study

There is a need for a treatment for colds due to EV/RV infection that could reduce the duration of symptoms and potentially the risk of complications. This study will evaluate the safety and efficacy of NTZ in the treatment of colds due to EV/RV infection.

#### 3. STUDY OBJECTIVES

Primary Objective: To evaluate the effect of NTZ in reducing the time to Sustained

Response compared to placebo in subjects with laboratory-confirmed

EV/RV infection

Secondary Objective: To evaluate the proportion of subjects requiring systemic antibiotics for

an infection secondary to EV/RV, including pneumonia, otitis media,

bronchitis, sinusitis or pharyngitis

Exploratory Objectives: i. To evaluate the proportion of subjects positive for EV/RV by PCR

at each of Days 4 and 10

ii. To evaluate the proportion of subjects requiring systemic antibiotics for any and each infection secondary to EV/RV, including

pneumonia, otitis media, bronchitis, sinusitis or pharyngitis

Safety Objective: To evaluate safety by analysis of adverse events

#### 4. STUDY DESIGN

# 4.1. Study Design Overview

This study is a multicenter, randomized, double-blind, placebo-controlled trial designed to evaluate efficacy and safety of NTZ 600 mg administered orally twice daily for five days compared to a placebo for the treatment of colds due to EV/RV infection.

18

Subjects will be stratified according to the following criteria:

Severity of Illness:

- <u>Mild illness</u> defined as baseline assessments of (1) at least one respiratory domain\* with a baseline score ≥2 <u>and</u> (2) resting pulse <90 beats per minute <u>and</u> (3) resting respiratory rate <20 breaths per minute.
- Moderate illness defined as baseline assessments of

   (1) at least one respiratory domain\* with a baseline score ≥2 and either (2) resting pulse ≥90 beats per

minute or (3) resting respiratory rate  $\geq$ 20 breaths per minute.

\* For this purpose, respiratory domains shall include the following 5 FLU-PRO domains/subdomains: chest, cough, nose, throat and head.

Time from onset of symptoms to randomization:

Risk of severe illness (per CDC):

<36 hours/>36 hours

- At Increased Risk: Subjects with COPD, Type 2 diabetes mellitus, obesity (BMI≥30), chronic kidney disease, sickle cell disease, serious heart conditions (such as heart failure, coronary artery disease, or cardiomyopathies), asthma (moderate or severe), cerebrovascular disease, cystic fibrosis, hypertension or high blood pressure, immunocompromised state (due to immune deficiencies, HIV, use of corticosteroids, or use of other immune-weakening medications), neurologic conditions (e.g., dementia), liver disease, pulmonary fibrosis, past or present history of smoking, thalassemia, or type 1 diabetes mellitus. Subjects who are ≥65 years of age.
- Not At Increased Risk: Subjects with none of the above conditions

Within strata, subjects will be randomized 1:1 to one of the following groups:

- Group 1 (NTZ): Two NTZ 300 mg tablets b.i.d. for 5 days
- Group 2 (Placebo): Two placebo tablets b.i.d. for 5 days

The study is expected to take place from July 2020 through May 2021.

Data for subjects enrolled in concurrent study RM08-3008 (COVID-19 treatment study with the same selection criteria and procedures) with laboratory confirmed EV/RV infection at baseline will be allocated to this study for analysis and will count toward the 350 to 400 required subjects.

# 4.2. Rationale for Important Issues in the Study Design

#### 4.2.1. Choice of NTZ Dose and Duration of Treatment

The dose of NTZ used for this clinical trial (600 mg b.i.d. for 5 days) has been associated with reductions in durations of illness in subjects infected with influenza, EV/RV, and coronavirus. Dose-range-finding study RM08-3001 in subjects with influenza infection demonstrated a dose-dependent efficacy response with a 300 mg b.i.d. group demonstrating a non-significant improvement over placebo.

In clinical trials involving 2,659 subjects, adverse events reported by subjects receiving 600 mg NTZ b.i.d. for 5 days were similar to those of subjects receiving the placebo, with the exception of a higher rate of chromaturia (10.8% compared to 0.8% for the placebo). Studies of NTZ at

higher doses have shown dose-dependent increases in the frequency of reported diarrhea and other gastrointestinal side effects, therefore no higher dose is planned for this study.

#### 4.2.2. Choice of Control Group

A placebo control is appropriate for the study due to lack of any approved active control.

#### 4.2.3. Choice of Patient Population

The population to be studied includes adults and adolescents with colds consistent with EV/RV infection. Because there are no approved antivirals for the treatment of EV/RV, subjects will not be prevented from being prescribed rescue medication for complications if warranted. Therefore, participation in the study will not pose unreasonable risk to any eligible subject. Discussion of specific eligibility criteria is presented below.

#### 4.2.3.1. Choice of Signs and Symptoms Required for Inclusion

Data from studies RM08-3004 and RM08-3005 indicate that, in subjects infected with influenza, EV/RV or seasonal coronavirus, subjects with low symptom scores for the head, throat, nose, chest and cough symptom domains in the absence of elevated pulse or respiratory rate, illness may be expected to resolve quickly. These subjects have less opportunity to benefit from antiviral treatment. Further, subjects who indicate that symptoms are already improving are also unlikely to benefit from treatment. Therefore, subjects will be required to have a score  $\geq 2$  for two respiratory symptom domains (head, throat, nose, chest, or cough) or a score  $\geq 2$  for one respiratory symptom domain in the presence of elevated vital signs (pulse  $\geq 90$  beats per minute or respiratory rate  $\geq 16$  breaths per minute). Subjects will be excluded if they report having no symptoms (global assessment), being at their usual health, that their symptoms do not interfere with their usual activities, or that their symptoms have improved since yesterday. Subjects presenting with signs or symptoms consistent with severe COVID-19 (resting shortness of breath, resting pulse  $\geq 125$ , resting respiratory rate  $\geq 30$ ) will also be excluded from the study.

#### 4.2.3.2. Inclusion of Subjects At Least 12 Years of Age (No Upper Age Limit)

The population to be studied includes adults and adolescents at least 12 years of age with colds consistent with EV/RV infection. This is a population similar to those selected for studies RM08-3001, RM08-3002, RM08-3003, RM08-3004 and RM08-3005 of the NTZ 300 mg extended release tablets in more than 5,000 subjects with colds or influenza-like illness. No safety concerns have been identified from these clinical trials. Data from pharmacokinetics studies in healthy volunteers 12 to 17 years of age or 18 to 65 years of age indicate that the pharmacokinetics of the major NTZ metabolites, tizoxanide and tizoxanide glucuronide, following oral administration of a NTZ 500 mg tablet are similar for these age groups. Safety data is also similar for these age groups. Therefore, the adult dose is deemed appropriate for pediatric patients down to 12 years of age. Informed consent will be required for subject participation in this study (see Section 8.1.1). A signed assent form will be required for any minors enrolled (≤ 18 years of age or as local regulations apply) as well as signed parental/legal guardian consent by their parent/legal guardian allowing for the minor's participation.

#### 4.2.3.3. Inclusion of Subjects with Underlying Conditions

For the present study, some subjects (e.g., subjects >65 years of age, underlying asthma or COPD, diabetes mellitus, underlying cardiovascular disease, etc. – see Inclusion/Exclusion criteria) who are at higher risk of complications or exacerbations of underlying conditions will be allowed to participate if, in the judgment of the investigator, they are able to comply with protocol requirements and are not expected to require hospitalization. There is no approved antiviral for colds due to EV/RV, and subjects will not be prevented from being prescribed rescue medication for complications. Therefore, participation in the study will not pose unreasonable risk to any eligible subject.

The pharmacokinetics of the proposed dose of NTZ have been studied in subjects with renal and hepatic impairment and no dose adjustment is recommended in these populations. A thorough QTc study of NTZ at doses of 675 mg and 2700 mg found no prolongation of the QTc interval.

CYP450 inhibition assays indicate that tizoxanide inhibits CYP2C8 with an IC50 of  $4.3\mu M$ , but a mechanistic static model used for potential drug-drug interactions indicated that a clinical interaction stemming from CYP2C8 inhibition by tizoxanide is unlikely.

While tizoxanide is more than 99.9% bound to plasma proteins, an *in vivo* drug-drug interaction study found no interaction between NTZ and warfarin. Tizoxanide inhibits the BCRP transporter and therefore may affect the pharmacokinetics of BCRP substrates, such as rosuvastatin. Coadministration of NTZ and rosuvastatin for seven days led to a 40% increase in the  $C_{max}$  of rosuvastatin and 80% and 70% increases of rosuvastatin AUC<sub>0-t</sub> and AUC<sub>0- $\infty$ </sub>, respectively. However, the short duration of treatment in this study is not anticipated to cause adverse effects related to co-administration of NTZ and rosuvastatin.

For more detailed information, refer to the NT-300 Investigator's Brochure-COVID/VRI.

#### 4.2.3.4. Exclusion of Subjects with Significant Immunodeficiency

Individuals with significant immunodeficiency, such as patients undergoing chemotherapy, transplant recipients receiving immunosuppressive therapy, and HIV patients with very low CD4 counts are more susceptible to longer durations of illness and more likely to experience complications due to viral respiratory infections. This is an important population in which to study antiviral drugs for the treatment of viral respiratory infections. Nonetheless, these subjects will be excluded from the present study due to (1) the likelihood of longer viral shedding necessitating longer courses or higher doses of treatment than what is proposed in this study, and (2) the likelihood that symptoms of illness may present differently in immunocompromised persons compared to immunocompetent persons due to reduced ability to produce the immune response that results in symptoms (van der Vries et al. 2013, St. Jude Children's Research Hospital).

#### 4.2.4. Use of Vitamin B Complex Supplement

All subjects will receive a vitamin B complex supplement ( , , , ) one tablet twice a day with study medication. This dose follows the manufacturer's labeled dosing. The purpose of the supplement is to help mask any chromaturia attributed to NTZ and aid in maintaining study blinding. The supplement will supply each subject with the following Percent Daily Values based on a 2,000 calorie diet: vitamin B1 1,333%, vitamin B2 824%, vitamin B3 240%, vitamin B5 360%, vitamin B6 1000%, vitamin B7

100%, vitamin B12 15,000%, folate 100%, and vitamin C 267%. Considering this supplement will provide well beyond the needed daily allowance of these water-soluble vitamins, excess amounts are expected to be excreted in the urine and provide discoloration.

#### 4.2.5. Choice of Patient-Reported Outcome Instrument

This clinical trial will use the InFLUenza Patient-Reported Outcome Questionnaire (FLU-PRO).

FLU-PRO was developed with the support of the U.S. Department of Health and Human Services through the National Cancer Institute and the National Institutes of Allergy and Infectious Diseases, National Institutes of Health, in response to the need for improved metrics to evaluate treatment effect in clinical trials of drugs for the treatment of influenza and other respiratory tract viral diseases. It was developed and validated in accordance with FDA's guidance, "Patient-Reported Outcome Measures: Use in Medical Product Development to Support Labeling Claims." It has also been validated for use on an electronic device as part of an electronic diary ("eDiary") that can time stamp diary entries to ensure timely recording, thereby mitigating risks of recall bias. We will use an electronic diary for this clinical trial. FLU-PRO was separately validated for use in a population with non-influenza like illness and also has recently been used in vaccine studies with older adults for the prevention of RSV (Powers et al. 2018, Yu et al. 2020). Data from Romark studies RM08-3004 and RM08-3005 also indicates validity and ability to detect change in patients infected with *Enterovirus/Rhinovirus* or seasonal coronavirus.

#### 4.2.6. Choice of Primary Endpoint

The primary endpoint was developed using data collected from 1,467 subjects infected with influenza, *Enterovirus/Rhinovirus* or seasonal coronaviruses during Romark studies RM08-3004 and RM08-3005. The endpoint defines a level of symptom improvement that constitutes a meaningful within-patient change in health status. The determination of meaningfulness was based on empiric evidence derived from the use of anchor questions. The endpoint requires (1) oral temperature <100.4 °F, (2) reduction of total symptom severity score from the previous day, (3) the patient to provide confirmation that symptoms are at least somewhat better, and (4) no symptom domain increase except below background levels for the remainder of the study (sustained response). These background levels were derived based on symptom scores reported by patients at the time they also reported being at usual health.

#### 5. STUDY POPULATION

#### 5.1. Inclusion Criteria

- 1. Male or female outpatients at least 12 years of age
- 2. Presence of clinical signs and/or symptoms consistent with worsening or stable cold due to EV/RV infection (one of the following is required):
  - a. Presence of at least two respiratory symptom domains (head, throat, nose, chest, cough) with a score of  $\geq 2$  as determined by Screening FLU-PRO <u>OR</u>
  - b. Presence of at least one respiratory symptom domain (head, throat, nose, chest, cough) with a score of  $\geq 2$  as determined by Screening FLU-PRO with pulse rate  $\geq 90 \text{ OR}$

c. Presence of at least one respiratory symptom domain (head, throat, nose, chest, cough) with a score of ≥2 as determined by Screening FLU-PRO with respiratory rate ≥16

<u>AND</u> patient reported assessment that symptoms are present, the symptoms are not consistent with the subject's usual health, the symptoms interfere with daily activities, and the symptoms have worsened or remained the same relative to the previous day, as confirmed by responses to questions in the Screening FLU-PRO.

- 3. Onset of symptoms no more than 72 hours before enrollment in the trial. Onset of symptoms is defined as the earlier of the first time at which the subject experienced subjective fever or any respiratory symptom (head, throat, nose, chest, or cough symptoms).
- 4. Willing and able to provide written informed consent (including assent by legal guardian if under 18 years of age) and comply with the requirements of the protocol, including completion of the subject diary and all protocol procedures.

#### 5.2. Exclusion Criteria

- 1. [Criterion removed in protocol version 2.0 See Revision History in Appendix 1.]
- 2. Subjects who experienced a previous episode of acute upper respiratory tract infection, otitis, bronchitis or sinusitis or received antibiotics for these conditions within two weeks prior to and including study day 1.
- 3. Severely immunodeficient persons including:
  - Subjects with immunologic disorders or receiving immunosuppressive therapy (e.g., for organ or bone marrow transplants, immunomodulatory therapies for certain autoimmune diseases)
  - b. Subjects with untreated HIV infection or treated HIV infection with a CD4 count below 350 cells/mm<sup>3</sup> in the last six months
  - c. Subjects actively undergoing systemic chemotherapy or radiotherapy treatment for malignancy
  - d. Subjects using steroids as maintenance therapy for chronic conditions
- 4. Subjects with active respiratory allergies or subjects expected to require anti-allergy medications during the study period for respiratory allergies.
- 5. Females of childbearing potential who are either pregnant or sexually active without the use of birth control. Female subjects of child-bearing potential that are sexually active must have a negative baseline pregnancy test and must agree to continue an acceptable method of birth control for the duration of the study and for 1 month post-treatment. A double barrier method, oral birth control pills administered for at least 2 monthly cycles prior to study drug administration, an IUD, or medroxyprogesterone acetate administered intramuscularly for a minimum of one month prior to study drug administration are acceptable methods of birth control for inclusion into the study. Female subjects are considered of childbearing potential unless they are postmenopausal (absence of menstrual bleeding for 1 year or 6 months if laboratory confirmation of hormonal status), or have had a hysterectomy, bilateral tubular ligation or bilateral oophorectomy.
- 6. Subjects residing in the same household with another subject participating in the study.

- 7. Treatment with any investigational drug or vaccine therapy within 30 days prior to screening and willing to avoid them during the course of the study.
- 8. Receipt of any dose of NTZ within seven days prior to screening.
- 9. Known sensitivity to NTZ or any of the excipients comprising the study medications
- 10. Subjects unable to swallow oral tablets or capsules.
- 11. Subjects with known severe heart, lung, neurological or other systemic disease that the Investigator believes could preclude safe participation.
- 12. Subjects likely or expected to require hospitalization unrelated to cold during the study period.
- 13. Subjects who, in the judgment of the Investigator, will be unlikely to comply with the requirements of this protocol including completion of the subject diary.
- 14. Subjects taking medications considered to be major CYP2C8 substrates. Refer to Table 6 in Section 6.5.
- 15. Persons with any clinical sign or symptoms suggestive of severe systemic illness with COVID-19, including the following:
  - a. shortness of breath at rest,
  - b. resting pulse  $\geq 125$  beats per minute,
  - c. resting respiratory rate ≥30 breaths per minute, or
  - d. SpO<sub>2</sub>  $\leq$  93% on room air at sea level.
- 16. Subjects known to have a diagnostic test positive for SARS-CoV-2 or influenza infection within the preceding three weeks.

# 5.3. Study Population Diversity

The Sponsor will select clinical sites to support recruitment of a diverse and representative population, including older individuals and racial and ethnic minorities.

#### 6. STUDY INTERVENTION

# 6.1. Study Intervention(s) Administration

#### **6.1.1.** Study Intervention Description

NTZ 300 mg extended release tablets for use in this study are yellow, round, convex, film-coated, bi-layer tablets for oral administration. Each tablet contains 300 mg of NTZ and the inactive ingredients.

Placebo tablets will have the same appearance and inactive ingredients as the active NTZ 300 mg extended release tablet.

The vitamin B complex supplement is manufactured by

The supplement will supply each subject with the following Percent Daily Values based on a 2,000-calorie diet: vitamin B1 1,333%, vitamin B2 824%, vitamin B3

240%, vitamin B5 360%, vitamin B6 1000%, vitamin B7 100%, vitamin B12 15,000%, folate 100%, and vitamin C 267%.

#### 6.1.2. Dosing and Administration



The food prior to drug intake should preferably be a high-fat meal, but at minimum a cereal bar.

All subjects will receive a vitamin B complex supplement one tablet twice a day (manufacturer's labeled dosing) to help mask any potential chromaturia attributed to NTZ and aid in maintaining study blinding.

# 6.2. Preparation, Handling, Storage and Accountability

#### 6.2.1. Acquisition and Accountability

Study medication will be provided by the Sponsor to the Investigational Site for dispensing.

Drug accountability will be tracked using an IWRS/IRT system as described in the study-specific Data Management Plan. Unused supplies must be returned to the Sponsor or destroyed in accordance with institutional procedures in effect at the study Site.

#### 6.2.2. Packaging and Labeling

NTZ or placebo tablets will be packaged in white 30 cc HDPE bottles, each containing 20 tablets. The kits will be stored at room temperature and will bear labels with the following information:

Table 5: Investigational Medication Label

20 Tablets Study No. RM08-3009 Treatment No: XXXX

Lot No: XXXX

Take 2 Tablets by Mouth with Food Twice Daily

Caution: New Drug – Limited by Federal Law to Investigational Use

STORE AT ROOM TEMPERATURE • DO NOT USE BEYOND END OF STUDY

KEEP OUT OF REACH OF CHILDREN

Study Sponsor: The Romark Institute for Medical Research

3000 Bayport Drive, Suite 200, Tampa, FL 33607

# 6.3. Randomization and Blinding

Subjects will be randomized 1:1 to receive either NTZ + vitamin B complex or placebo + vitamin B complex. An independent third party will prepare a master randomization list and maintain the masking of the study. Subjects who qualify for the study will be assigned to treatment using centralized randomization procedures. The treatment numbers will appear on the bottles containing the masked study medication. The randomization list will be masked to study participants including Sponsor, Investigators, study monitors, statisticians, subjects and laboratory personnel. Unmasking procedures will be detailed in the Medical Monitoring Plan and Investigators will be provided instructions for unmasking.

# 6.4. Study Intervention Compliance

Subject compliance with study medication will be checked by site staff daily during the treatment period. Subjects will return the treatment kit with any unused medication to the clinic at the Day 10 visit. Subjects will be considered non-compliant (major protocol deviation) if they have missed more than two doses of the investigational medication during the first three days of the study. Non-compliance will not be cause for discontinuation of subject participation in the study.

# 6.5. Concomitant Therapy

The following medications will not be allowed during the study: topical or systemic decongestants, nasal corticosteroids, and any prescription or non-prescription medications classified as (i) expectorants and cough preparations, (ii) analgesics and antipyretics, (iii) antihistamines (American Hospital Formulary Service (AHFS) classification) or (iv) medications considered major CYP2C8 substrates (see Table 6 below). As an exception to this rule, subjects will be allowed to use acetaminophen and/or dextromethorphan as necessary for disabling symptoms.

**Table 6:** Major CYP2C8 Substrates

| Generic Name | Brand Name(s) | Therapeutic Use and/or Drug Class |
|---|---|---|
| Amodiaquine | BASOQUIN, CAMOQUIN,<br>FLAVOQUIN | Antimalarial |
| Daprodustat (GSK1278863) | * | Antianemic, prolyl hydroxylase inhibitor |
| Dasabuvir (ABT-333) | EXVIERA | Antiviral, NSB5 inhibitor |
| Enzalutamide | XTANDI | Anticancer, antiandrogen |
| Montelukast | SINGULAIR | Antiasthmatic, LTRA |
| Pioglitazone | ACTOS | Antidiabetic, PPAR-γ agonist |
| Repaglinide | NOVONORM, PRANDIN | Antidiabetic, meglitinide analog |

Source: Backman et al. 2016

Subjects are also prohibited from taking hydroxychloroquine, chloroquine, remdesivir, azithromycin or lopinavir/ritonavir during the study except as standard-of-care rescue medication.

<sup>\*</sup>Currently listed as investigational only and not yet granted a trade name by the manufacturer

Medications for pre-existing conditions that are not excluded (see exclusion criteria) should be continued as prescribed. Standard-of-care rescue medication is permitted for complications of COVID-19 illness. The use of such medication will be recorded in the EDC system.

# 7. STUDY INTERVENTION DISCONTINUATION AND PARTICIPANT DISCONTINUATION

Treatment will be discontinued for individual subjects for the following reasons:

- 1. An allergic reaction occurs or is suspected.
- 2. Medical conditions that may require investigational medication discontinuation in the Investigator's judgment.
- 3. Subject desire to discontinue participation.

In the case of an allergic reaction or other medical condition requiring subject discontinuation, appropriate treatment will be instituted by the Investigator.

Subjects will be encouraged to complete all protocol-specified follow-up visits even if study drug is withdrawn.

#### 8. STUDY PROCEDURES

#### 8.1. Visit Procedures

Study procedures to be completed at each visit are indicated in the Schedule of Assessments. Descriptions of selected procedures are outlined in the following sections.

#### 8.1.1. Informed Consent

Each subject must give written consent according to local requirements after the nature of the study has been fully explained. The informed consent form (ICF) must be signed before performance of any study-related activity. The informed consent form will be approved by both the Sponsor and by the reviewing IRB. They will be in accordance with principles that originated in the Declaration of Helsinki, current ICH and GCP guidelines, applicable regulatory requirements, and Sponsor policy. The ICF may be signed using wet ink or digital signature.

Before enrollment in the study, the Investigator or an authorized member of the investigational staff must explain to potential subjects the aims, methods, reasonably anticipated benefits, and potential hazards of the study, and any discomfort participation in the study may entail. Subjects will be informed that their participation is voluntary and that they may withdraw consent to participate at any time. They will be informed that choosing not to participate will not affect the care he/she will receive. Finally, they will be told that the Investigator will maintain a subject identification register for the purposes of long-term follow-up if needed and that their records may be accessed by health authorities and authorized Sponsor staff without violating the confidentiality of the subject, to the extent permitted by the applicable law(s) or regulations. By signing the ICF the subject is authorizing such access, and agrees to allow his or her study physician to re-contact the subject for the purpose of obtaining consent for additional safety evaluations, if needed. Only

subjects who are fully able to understand the risks, benefits, and potential AEs of the study, and provide their consent voluntarily will be enrolled.

The subject will be given sufficient time to read the ICF and the opportunity to ask questions. After this explanation and before entry into the study, consent should be appropriately recorded by means of the subject's personally dated signature. After having obtained the consent, a copy of the ICF must be given to the subject.

If the subject is unable to read or write, an impartial witness should be present for the entire informed consent process (which includes reading and explaining all written information) and should personally date and sign the ICF after the oral consent of the subject is obtained, if permitted by local law.

Assent from any minor ( $\leq$  18 years of age or as local regulations apply) enrolled into the study will be obtained along with documented consent from their parent/legal guardian to allow the minor to participate in the study. The assent and consent forms must be signed prior to the performance of any study related activity.

Signed ICFs must remain in the subject's file(s) and be available for verification by representatives of Romark, the IRB, and FDA/relevant regulatory agencies at any time.

#### 8.1.2. Medical History

All relevant medical history should be entered in the EDC system at the Screening visit. Relevant medical history includes:

- 1. Any disease, condition or surgery active at the time of the Screening visit;
- 2. Any disease, condition or surgery ending within two months of the Screening visit; or
- 3. Any other disease, condition or surgery relevant to the subject's infection or clinical management.

#### 8.1.3. Physical Examination

Physical examinations will include assessment of each body system including skin, head (eye, ear and nose), neck, mouth/throat, lymph nodes, cardiovascular, respiratory, gastrointestinal, neurological, and musculoskeletal systems as well as general appearance for abnormalities.

The Investigator will complete a full physical examination at the Screening visit. Physical examinations should occur at follow-up and unscheduled visits as required by symptoms or adverse changes from baseline.

### 8.1.4. Body Measurements and Resting Vital Signs

Body measurements and resting vital signs will include assessment of the following:

- 1. Height (Screening visit only)
- 2. Weight
- 3. Oral temperature
- 4. Blood pressure

- 5. Pulse rate
- 6. Respiratory rate
- 7. Oxygen saturation

#### 8.1.5. Screening FLU-PRO

The FLU-PRO questionnaire will be administered during the Screening visit to confirm symptoms required for eligibility.

#### 8.1.6. Randomization and Dispensing Study Medication

Randomization and study medication kit assignment will be accomplished using an Interactive Randomization Tool (IRT) feature in the EDC system after all screening procedures have been completed and the subject has been determined to be eligible for the study. Site staff will witness the subject take the first dose of study medication in the clinic as soon as possible following randomization and record the date and time of medication intake in the EDC system.

#### 8.1.7. Subject Instructions

At each subject contact, site staff will instruct the subject regarding:

- Administration of study medication. Subjects will be instructed to take the study medication (two tablets) twice daily with the morning and evening meals, approximately every 12 hours (< 1 hour after food intake, preferably a high-fat meal but at a minimum a cereal bar) and a B complex vitamin
- 2. Completion of subject diary. Subjects will be reminded to complete the electronic diary and any questions will be answered.
- 3. Use of birth control. Female subjects of childbearing potential, if sexually active, will be instructed to continue an acceptable method of birth control for the duration of the study and for 1 month post-treatment. Acceptable methods of birth control include a double barrier method, oral birth control pills, an IUD, or medroxyprogesterone acetate administered intramuscularly.
- 4. *Follow-up visits*. Subjects will be reminded of the study schedule and of the next scheduled visit.
- 5. Seeking emergency care or contacting the study physician or nurse. Subjects must be informed to seek emergency medical care or contact the study physician or nurse if they develop any of the following symptoms listed below at any point during the study.

#### **CONTACT STUDY PHYSICIAN IF YOU HAVE:**

- Trouble breathing including shortness of breath
- Severe headache, stiff neck, confusion or excessive somnolence
- If fever ( $\geq$ 99°F or  $\geq$ 37.2°C) returns after being absent for 24 hours
- · Increased difficulty breathing

- Wheezing develops
- New pain develops or pain localizes to one area, such as an ear, the throat, the chest, or the sinuses
- Symptoms become more severe or frequent
- Symptoms recur or any difficulty breathing following 5-10 days resolution of illness
- An allergic-like reaction occurs or is suspected
- Abnormal behavior

# 8.1.8. Day 2-7 Subject Contact

Site staff will contact each subject by telephone on study Days 2-7 to verify:

- 1. Did the subject take all expected doses of study medication?
- 2. Did the subject complete all expected electronic diaries?
- 3. Does the subject have worsening symptoms or adverse events that warrant an unscheduled visit?
- 4. Does the subject have shortness of breath at rest? If yes, instruct the subject to come to the clinic for an unscheduled visit to screen for progression of illness or refer to hospital as warranted. If the subject is referred to the hospital or emergency department, the Investigator will attempt to obtain hospital records indicating SpO<sub>2</sub> or PaO<sub>2</sub>/FiO<sub>2</sub> from the subject for the purposes of defining progression to severe COVID-19 illness. The SpO<sub>2</sub> or PaO<sub>2</sub>/FiO<sub>2</sub> obtained from hospital records will be entered on an Unscheduled Visit eCRF.

If the subject has missed medication or electronic diaries, the site staff will re-train the subject on the importance of medication and diary compliance.

This contact may occur at the Day 4 or unscheduled visit in lieu of telephone contact.

#### 8.1.9. Day 28 Subject Contact

Site staff will contact each subject by telephone on study Day 28 to determine if the subject has experienced any new adverse events, developed severe COVID-19 illness, or required hospitalization for any reason.

If warranted, the Day 28 subject contact may also occur in-person at the clinic or another location as agreed upon by the site and subject.

# 8.2. Laboratory Assessments

#### 8.2.1. Assessments in the Clinic

A urine pregnancy test will be performed in the clinic only for women of childbearing potential (post-menarche, pre-menopause, not surgically sterile) at the Screening visit.

#### 8.2.2. Central Laboratory Assessments

A central laboratory will be used for safety and diagnostic virology testing. A laboratory manual will be provided to each clinical site with sample collection and handling details.

#### 8.2.2.1. Laboratory Safety Assessments

Blood tests for safety monitoring will include hemoglobin, hematocrit, complete blood count (total and differential), platelet count, random blood sugar, total cholesterol, HDL, LDL, triglycerides, albumin, AST, ALT, GGT, alkaline phosphatase, bilirubin (total/direct), BUN, creatinine, sodium, potassium, chloride.

Routine urinalysis will include appearance, glucose, protein, and blood.

#### 8.2.2.2. Diagnostic Virology Testing

Diagnostic virology testing will be performed using nasopharyngeal swab samples collected at the Baseline, Day 4 and Day 10. The nasopharyngeal sample for virology testing will be collected using a single nasopharyngeal swab inserted into both nostrils in accordance with procedures detailed in the study-specific laboratory manual.

The ePlex® Respiratory Pathogen Panel (GenMark, Carlsbad, CA) will be used to detect influenza A (non-specific as to subtype); influenza A H1, H1N1 (2009), H3 subtypes; influenza B; RSV A and B; parainfluenza 1, 2, 3 and 4; hMPV; adenovirus; human EV/RV; coronavirus NL63, HKU1, 229E and OC43; Chlamydophila pneumoniae; and Mycoplasma pneumoniae.

The Aptima® SARS-CoV-2 Assay (Hologic, Inc, San Diego, CA) will be used to detect SARS-CoV-2.

All Baseline nasopharyngeal swabs will be tested by both PCR assays.

Post-baseline samples (Days 4 and 10) will only be tested by the ePlex Respiratory Pathogen Panel (RPP) and will only be tested if the sample from the preceding timepoint was positive for EV/RV. For example, a subject who is positive for EV/RV at Baseline will have the Day 4 sample tested by the ePlex RPP. If the subject's Day 4 sample is negative for EV/RV, the Day 10 sample will not be tested.

#### 8.2.3. Pharmacokinetics Assessments

Blood samples for pharmacokinetics analysis will be sent to the central laboratory by the site and shipped to a referral laboratory for analysis. Sample collection and handling details will be included in the central laboratory manual.

#### 8.2.4. Plan for Monitoring Viral Resistance

If any Day 10 nasopharyngeal swab sample is positive for EV/RV by the ePlex RPP, the Baseline and Day 10 nasopharyngeal swab samples for the subject will be tested for post-treatment reduced susceptibility to tizoxanide.

#### 8.3. Subject Diary

The subject diary will be used to generate primary efficacy data. Therefore, diary compliance is of critical importance.

#### 8.3.1. Subject Diary Completion

Subjects will complete a diary including:

- Oral temperature taken using the study thermometer twice daily (morning and evening),
   and
- The FLU-PRO© symptoms questionnaire daily in the evening.

The diary will be completed using the subject's smartphone or provisioned device.

Site staff will ensure subject access and ability to complete the diary during the Baseline visit by having the subject complete a practice diary in the office. Subjects will complete the first post-Screening diary at home on the evening of study Day 1.

Subjects will receive electronic reminders to complete the diary daily to ensure compliance.

#### 8.3.2. Subject Diary Compliance Monitoring

It is the responsibility of the clinical site to ensure that subjects are completing the diary as directed. E-mail notifications will be sent to the site daily with a list of subjects who missed the previous day's diary in order to direct follow-up contact with the subject to re-train on the importance of the diary. Site staff may also view a diary completion report at any time within the EDC system.

#### 8.4. Adverse Events and Serious Adverse Events

#### 8.4.1. Definitions

The following definitions will apply to the reporting of adverse events:

- 1. Adverse Event: Any unwanted physical, psychological or behavioral change experienced by a subject during the course of the study and after taking the first dose of study medication regardless of its severity or relation to the study. Adverse events may include symptoms, signs, unexpected worsening of pre-existing conditions, clinically significant changes in laboratory values, diseases and syndromes, and significant and unexpected failures of pharmacological action of other medications. Symptoms of viral respiratory infections (VRIs) (cough, sore, throat, nasal obstruction, fatigue, headache, myalgia, or feverishness) will not be reported as adverse events.
- 2. Serious Adverse Event: Any adverse experience occurring at any dose that is fatal or life threatening; requires in-patient hospitalization or prolongation of an existing hospitalization; is a persistent significant disability/incapacity; is a congenital anomaly or birth defect; or is an important medical event that may not result in death, be life-threatening, or require hospitalization but, based upon appropriate medical judgment, may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed above.
- 3. <u>Unexpected Adverse Event:</u> Any adverse experience that is not identified in nature, severity, or frequency in the Investigator's Brochure for NTZ.
- 4. <u>Severity of adverse events</u> will be assessed as mild, moderate, severe or potentially life-threatening by the Investigator using the Toxicity Grading Scale Tables provided in Appendix 4 (derived and adapted from "Guidance for Industry: Toxicity Grading Scale for

Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials", US Dept. of HHS, FDA, CDER, September 2007 and the National Institutes of Health, National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0).

#### 5. Causality (relationship to treatment) will be assessed as follows:

- Definitely Related: The adverse event is clearly related to the investigational agent(s) or research intervention: the adverse event has a temporal relationship to the administration of the investigational agent(s) or research intervention, follows a known pattern of response, and no alternative cause is present.
- Probably Related: The adverse event is likely related to the investigational agent(s) or intervention: the adverse event has a temporal relationship to the administration of the investigational agent(s) or research intervention, follows a known or suspected pattern of response, but an alternative cause may be present.
- Possibly Related: There is a reasonable possibility that the event may have been
  caused by or is linked in a significant way to the research; the adverse event has a
  temporal relationship to the administration of the investigational agent(s) or research
  intervention, follows a suspected pattern of response, but an alternative cause is
  present.
- *Unrelated (or Not Related)*: The adverse event is clearly NOT related to the investigational agent(s) or intervention: the adverse event has no temporal relationship to the administration of the investigational agent(s) or research intervention, follows no known or suspected pattern of response, and an alternative cause is present.

Under double-blind treatment conditions, it should be assumed that all subjects are taking the test drug.

#### 8.4.2. Recording and Follow Up of Adverse Events

At the time of each visit, the subject will be questioned regarding the occurrence and nature of any adverse events and all events will be recorded in the subject's medical records and in the EDC system. Any subject affected will be examined by the Investigator as deemed necessary to ascertain the course of the event and any residual effects. All adverse events must be followed until their resolution or stabilization even beyond the planned study period.

All moderate and severe adverse events will be reviewed by the Principal Investigator who will determine using his/her best clinical judgment whether they warrant the subject to be discontinued from the study. The Sponsor will be notified immediately if a subject is discontinued from the study. For all adverse events that require the subject to be discontinued from the study, relevant clinical assessments and laboratory tests will be repeated as clinically indicated until final resolution or stabilization of the event(s).

All subjects will be instructed to contact the Investigator, Investigator's assistants, or clinical personnel should the subject have any serious adverse experiences.

An overdose is defined as any intentional or unintentional consumption of the drug by any route that exceeds the highest dose stated in the Investigator's Brochure or in an investigational protocol,

whichever dose is larger. Overdoses without an associated adverse event should be recorded, but not reported as an adverse event.

#### 8.4.3. Reporting Requirement

The Principal Investigator is required to notify The Romark Institute for Medical Research (Sponsor) immediately (within 24 hours of the initial report) of any unexpected, fatal, or life-threatening experience and all unusual, alarming, or serious reactions to medication regardless of any opinions as to the cause/effect relationship. All serious adverse events will also be reported to the IRB as required by the IRB procedures. Adverse events should be reported to:

The Romark Institute for Medical Research



#### 8.4.4. Medication Errors

A medication error is defined as any preventable event related to dosing instructions, product labeling, or packaging that causes or leads to inappropriate medication use or subject harm while the medication is in the control of the investigative site or subject. Medication errors which result in adverse events should be recorded and reported as adverse events. All other medication errors should be reported to the study Sponsor through the Medical Affairs department within 7 days of identification by the site.

#### 9. STATISTICAL CONSIDERATIONS

# 9.1. Sample Size Determination

The primary efficacy parameter is the time from first dose to Sustained Response based on the FLU-PRO Patient Reported Outcomes instrument (see Section 9.3). This response definition was applied to data from Romark study RM08-3005 in the treatment of colds caused by EV/RV. See Section 2.2.4 for the Kaplan-Meier curves forming the basis for sample size calculations for this study.

These assumptions yield a sample size of 312 subjects (156 per group). These calculations were performed for the Gehan rank test using SAS PROC POWER (SAS 9.4) with the curves shown in Section 2.2.4 (proportion not responded by the end of each day was used as input) and censoring at day 21. In order to ensure a robust dataset, we have selected a sample size of at least 350 subjects with laboratory-confirmed EV/RV infection including an allowance for approximately 10% of subjects to discontinue early or otherwise have missing data.

# 9.2. Efficacy Variables

Primary Efficacy Parameter: Time from first dose to Sustained Response based on the FLU-PRO Patient Reported Outcomes Instrument.

Secondary Efficacy Parameter: Proportions of subjects requiring systemic antibiotics for an

infection secondary to EV/RV, including pneumonia, otitis

media, bronchitis, sinusitis or pharyngitis

Exploratory Efficacy Parameters: i. Proportion of subjects positive for EV/RV by PCR at Days 4 and 10.

 ii. To evaluate the proportion of subjects requiring systemic antibiotics for any and each infection secondary to EV/RV, including pneumonia, otitis media, bronchitis, sinusitis or pharyngitis

# 9.3. Response Definitions

# 9.3.1. Response Definitions for the Primary Efficacy Analysis

Sustained Response:

A decrease in total FLU-PRO score from the previous diary with patient assessment that symptoms are at least "somewhat better than yesterday", no oral temperature ≥100.4°F in the prior 24 hours, and no future increase in any of the FLU-PRO domains except within the following levels:

| FLU-PRO Domain* | Background Level |
|------------------|---------------------------------------------------------|
| Body/Systemic | 0.56 |
| Throat | 0.67 |
| Eyes | 0.67 |
| Gastrointestinal | 2.00 |
| Head | 2.00 |
| Nose | Score at time of response or 0.75, whichever is greater |
| Chest | Score at time of response or 0.00, whichever is greater |
| Cough | Score at time of response or 1.75, whichever is greater |

<sup>\*</sup> A diagram of the FLU-PRO domain/subdomain structure is attached as Appendix 5.

Time of Sustained Response:

The time of the first diary at which all Sustained Response criteria are met.

Time to Sustained Response:

The time (hours) from the first dose of study medication and the Time of Sustained Response.

#### **9.3.2.** Definitions for Complications of Colds

Complications of colds are infections secondary to colds requiring systemic antibiotics, including pneumonia, otitis media, bronchitis, sinusitis and pharyngitis. Diagnostic criteria for these infections are as follows:

Bacterial Pneumonia (criteria from FDA Guidance for Industry, *Community-Acquired Bacterial Pneumonia: Developing Drugs for Treatment*):

- 1. At least two of the following symptoms: difficulty breathing, cough, production of purulent sputum, chest pain, and
- 2. At least two of the following vital sign abnormalities: fever, hypotension, tachycardia, tachypnea, and
- 3. At least on of the following findings: hypoxemia, clinical evidence of pulmonary consolidation, elevated white blood cell count or leukopenia, and
- 4. If performed, chest radiograph findings of new infiltrates in a lobar or multilobar distribution, and
- 5. If performed, microbiologic criteria: appropriate sputum specimen with fewer than 10 squamous epithelial cells and more than 25 polymorphonuclear cells per low power field.

Acute Bacterial Otitis Media (criteria from FDA Guidance for Industry, *Acute Bacterial Otitis Media: Developing Drugs for Treatment*):

- 1. Symptoms of ear pain or ear ache, ear fullness or decreased hearing, and
- 2. One or more of the following otoscopic findings performed by a clinician experienced in otoscopy:
  - a. Bulging or fullness of the tympanic membrane (convexity of the plane of the eardrum), with loss of anatomic landmarks on visualization,
  - b. Opacification of the tympanic membrane regardless of color,
  - c. Erythema of the tympanic membrane, or
  - d. If performed, abnormal tympanic membrane mobility on biphasic pneumatic otoscopy (a tympanic membrane in the neutral position or retracted is not sufficient evidence of acute bacterial otitis media because these findings are not specific enough to distinguish the disease from otitis media with effusion)

Acute Bacterial Sinusitis (criteria derived from FDA Guidance for Industry, *Acute Bacterial Sinusitis: Developing Drugs for Treatment*):

- 1. At least two of the following symptoms:
  - Maxillary tooth pain (unilateral findings can be more specific)
  - Facial pain (unilateral findings can be more specific)
- Frontal headache
- Purulent nasal discharge (unilateral findings can be more specific)
- New onset fetor oris (bad breath)
- Morning cough
- Nasal obstruction
- 2. At least one of the following signs:
  - Purulent secretions from sinus ostia on examination
  - Abnormal sinus transillumination
  - Pain on palpation over sinuses
  - Facial swelling
- 3. If performed, radiographic findings consistent with acute sinusitis

Acute Streptococcal Pharyngitis (criteria derived from IDSA, Clinical Practice Guideline for the Diagnosis and Management of Group A Streptococcal Pharyngitis):

- 1. Sore throat consistent with acute streptococcal pharyngitis and
- 2. Throat swab sample positive for group A streptococcus by rapid antigen detection test (RADT) and/or culture.

Acute Bacterial Bronchitis (criteria derived from FDA Guidance for Industry, *Acute Bacterial Exacerbations of Chronic Bronchitis in Patients with Chronic Obstructive Pulmonary Disease* and Knutson and Braun 2002):

- 1. New or increased cough, dyspnea or chest tightness
- 2. New or increased sputum production
- 3. Presence of tachypnea, wheezing, ronchi, crackles or prolonged expiration
- 4. History and physical examination rules out other causes of cough
- 5. No evidence of pulmonary consolidation

# 9.4. Statistical Methodology

The statistical methodology is described briefly below and will be described in detail in the Statistical Analysis Plan.

## 9.4.1. Efficacy Analyses

Efficacy analyses will be based on a population consisting of all subjects randomized who receive at least one dose of study medication and are positive for EV/RV by PCR at Baseline. For time-to-event analyses, a test of significance (as described in the following) will be performed with descriptive statistics provided, including the use of Kaplan-Meier figures.

There will be one primary efficacy analysis:

Time to Sustained Response for the NTZ treatment group will be compared to that of the
placebo treatment group using a stratified Gehan-Wilcoxon test (α=0.05) where
stratification will follow that used for randomization. Subjects without a Sustained
Response recorded will be treated as censored as of the last diary without a documented
Sustained Response.

If the primary analysis is significant at the 0.05 level, the key secondary efficacy analysis will be formally evaluated at the 0.05 level as follows:

Proportions of subjects requiring systemic antibiotics for an infection secondary to EV/RV, including pneumonia, otitis media, bronchitis, sinusitis or pharyngitis, will be compared between the treatment groups using a Cochran-Mantel-Haenszel (CMH) test stratified by the randomization strata. Note that the study is not powered to detect statistically significant differences for this analysis.

Exploratory analyses will be performed as follows:

- Proportions of subjects positive for EV/RV by PCR at study Day 4 and Day 10 will be compared between the treatment groups using a Cochran-Mantel-Haenszel (CMH) test stratified by the randomization strata.
- Proportions of subjects requiring systemic antibiotics for each of pneumonia, otitis media, bronchitis, sinusitis or pharyngitis, will be compared between the treatment groups using a Cochran-Mantel-Haenszel (CMH) test stratified by the randomization strata.

This trial is being conducted during the COVID-19 pandemic and is likely to enroll significant numbers of subjects with COVID-19. Prior to database lock and unblinding, a pooled analysis of the blinded subject data will be completed to count the number of subjects with laboratory-confirmed SARS-CoV-2 infection.

In the event that ≥350 subjects with laboratory-confirmed SARS-CoV-2 infection have been enrolled, it is expected that this will provide ≥90% power to detect a statistically significant difference in the Time to Sustained Response survival distributions between the NTZ and placebo treatment groups [two-sided alpha=0.05, calculations performed for the Gehan rank test using SAS PROC POWER (SAS 9.4) based upon data from Romark trials RM08-3004 and RM08-3005 assuming equal allocation of subjects across treatment arms]. In this case, subjects with laboratoryconfirmed SARS-CoV-2 will be analyzed under a separate Statistical Analysis Plan that will be signed and placed on file prior to database lock. The Statistical Analysis Plan will specify Time to Sustained Response (as described above) as the primary efficacy endpoint to be analyzed at the 0.05 level and a comparison of proportions experiencing progression to severe COVID-19 illness (defined as shortness of breath at rest and SpO<sub>2</sub> < 93% on room air) using a Cochran-Maentel-Haenszel (CMH) test stratified by the randomization strata as the key secondary analysis. Day 4 and Day 10 nasopharyngeal swabs will be analyzed for the presence of SARS-CoV-2 for all subjects positive for SARS-CoV-2 at Baseline and Day 22 nasopharyngeal swabs will be analyzed if the Day 10 sample is positive for SARS-CoV-2 [analysis using Aptima® SARS-CoV-2 Assay (Hologic, Inc, San Diego, CA) as described in Section 8.2.2.2]. Proportions of subjects positive for SARS-CoV-2 at Day 4 and Day 10 will be compared across treatment groups using a CMH test stratified by the randomization strata as an exploratory analysis. Serology samples will be analyzed for quantitative IgG and IgM antibodies and descriptive statistics of the results will be

presented by treatment group. Safety and pharmacokinetics will be analyzed as described in sections 9.4.2 and 9.4.3 below.

## 9.4.2. Population Pharmacokinetics Analysis

On Day 4, plasma samples will be collected before the morning dose (at the trough) for determination of drug concentration. These data will allow for analysis of relationships between trough plasma concentrations and clinical and virologic response.

Trough plasma concentrations of tizoxanide and tizoxanide glucuronide will be summarized descriptively for NTZ-treated subjects. Exploratory analyses will be conducted to evaluate the relationships between plasma concentrations and age, race, gender, body weight, body mass index, VRI and adverse events.

## 9.4.3. Safety Analyses

All randomized subjects who receive at least one dose of study medication will be evaluated for drug safety. Safety analyses will be done descriptively.

#### 10. OPERATIONAL CONSIDERATIONS

## 10.1. Regulatory, Ethical and Study Oversight Considerations

#### 10.1.1. Ethics

The clinical trial will be performed in accordance with the guidelines set by the World Medical Assembly (Declaration of Helsinki, last amendment in Fortaleza, Brazil, October 2013).

Informed consent will be obtained from each subject as described in Section 8.1.1.

Prior written approval of the study protocol and of the informed consent form will be obtained by the Sponsor from the appropriate central or local IRB.

Prior to study initiation, the Investigator will provide the IRB with required documents for review and approval. See Appendix 3: List of Essential Documents for designation of documents that may be required by the IRB prior to study initiation or during the course of study conduct. No site will screen subjects until the IRB has given full approval of required documents and the data approval letter identifying the IRB and the documents approved is delivered to the study Sponsor.

For all protocol amendments (excluding the ones that are purely administrative, with no consequences for subjects, data or study conduct), the amendment and applicable informed consent form and assent form revisions must be submitted promptly to the IRB for review and approval before implementation of the change(s), except when necessary to eliminate immediate hazard to the study subjects. If a deviation from, or a change to the protocol was implemented to eliminate an immediate hazard to study subjects, then the implemented deviation or change, the reasons for it, and, if appropriate, the protocol amendment should be submitted to the IRB as soon as possible.

The re-approval of the clinical study by the IRB should be documented in writing.

At the end of the study, the Investigator (or Sponsor where required) will notify the IRB about the study completion.

#### 10.1.2. Investigator Responsibilities

The Investigator is responsible for ensuring that the clinical study is performed in accordance with the protocol, current International Conference on Harmonization (ICH) guidelines on Good Clinical Practice (GCP), and applicable regulatory and country specific requirements.

Good Clinical Practice is an international ethical and scientific quality standard for designing, conducting, recording, and reporting studies that involve the participation of human subjects. Compliance with this standard provides public assurance that the rights, safety, and wellbeing of study subjects are protected, consistent with the principles that originated in the Declaration of Helsinki, and that the clinical study data are credible.

## 10.1.3. Quality Assurance and Quality Control

The accuracy and reliability of the study data will be assured by the selection of qualified Investigators and appropriate study centers, review of protocol procedures with the Investigator and associated personnel prior to the study, and by periodic monitoring visits by the Sponsor or Sponsor's representatives (see Section 10.1.6). Written instructions will be provided for collection, preparation and shipment of biological samples.

The Sponsor will be entitled to inspect and audit the facilities used in the clinical and laboratory parts of the study, as well as to make anonymized copies of all the data files pertaining to the study. Similar procedures may also be conducted by agents of any regulatory body, either as part of a national GCP compliance program or to review the results of this study in support of a regulatory submission. The Investigator should immediately notify the Sponsor if they have been contacted by a regulatory agency concerning an upcoming inspection.

Quality oversight of study management will be accomplished according to the study-specific Integrated Quality and Risk Management Plan.

#### 10.1.4. Safety Oversight

The Sponsor and Medical Monitor will be responsible for safety oversight of the study. Procedures for safety oversight are described in the study-specific Medical Monitoring Plan.

## 10.1.5. Data Handling and Record Keeping

#### 10.1.5.1. Data Collection and Management Responsibilities

Sponsor Data management will be responsible for oversight of data collection, cleaning and locking according to the study-specific Data Management Plan.

Data will be collected on site-specific source data forms and transcribed into an electronic data capture (EDC) system by site staff. The responsible study monitor(s) will verify data according to the Clinical Monitoring Plan, either remotely or at the clinical study site. The Investigator will ensure that the data recorded are accurate and complete.

Queries emerging during data cleaning will be generated within the EDC system by monitors or data management personnel. The Investigator and/or designee will answer the queries and update the source data, as needed.

#### 10.1.5.2. Study Records Retention

The Investigator/institution will maintain all CRFs, EDC source forms, and source documents that support the data collected from each subject, as well as all study documents as specified in ICH/GCP Section 8, and all study documents as specified by the applicable regulatory requirements for the duration required by applicable regulatory authorities or until the Sponsor informs the Investigator/institution that these documents are no longer needed.

If it becomes necessary for the Sponsor or the appropriate regulatory authority to review any documentation relating to this study, the Investigator must permit access to such reports.

The Sponsor will be responsible for maintaining the Trial Master File which is a clear documentation of the course of the study.

#### 10.1.6. Clinical Monitoring

Clinical monitoring will be conducted by the Sponsor and/or a contract research organization (CRO) according to the study-specific Clinical Monitoring Plan.

The Investigator will grant representatives of the Sponsor's clinical operations team and quality team, as well as regulatory agencies and ethical committees access to inspect facilities and records (including subject charts) relevant to this study and agrees to assist the monitors in their activities, if requested.

#### 10.1.7. Protocol Deviations

Protocol deviations will be documented by the Investigator, reported to the institutional review board (IRB) as appropriate, and also reviewed by the assigned clinical research associate. Deviations will be reported in the clinical trial management system or applicable EDC. Each deviation will be classified as major or minor according to the following definitions:

Major protocol deviation: A deviation that has an impact on subject safety, may substantially

alter risks to subjects, may have an effect on the integrity of the study data, or may affect the subject's willingness to participate in

the study

Minor protocol deviation: All other protocol deviations.

#### 10.1.8. Study Discontinuation and Closure

The study may be discontinued under the following circumstances:

- 1. The Sponsor reserves the right to discontinue the study at any time.
- 2. Adverse event listings will be produced for safety monitoring at least once every two weeks during recruitment. The data will be tested to determine if there are greater than 20% of the subjects who have had ≥ Grade 3 adverse events considered by the Investigator to be possibly, probably or definitely related to the study drug (defined by the Toxicity Grading Scale Tables provided in Appendix 4).

If greater than 20% of the subjects have at least one Grade 3 or Grade 4 adverse event considered to be possibly, probably or definitely related to the study drug by the study Medical Monitor, then the study must be stopped and the Institutional Review Boards, and

FDA's Division of Antiviral Drug Products will be notified. All safety and efficacy data will be submitted to the FDA in a timely manner.

#### 10.1.9. Data and Report Requirements

See Appendix 3: List of Essential Documents for designation of documents required from the Investigator by the Sponsor prior to approval and initiation of the study and before the study can be considered complete and terminated.

## 10.1.10. Confidentiality and Privacy

The collection and processing of personal data from subjects enrolled in this study will be limited to those data that are necessary to investigate the safety, quality, and utility of the investigational study drug(s) used in this study.

These data will be collected and processed with adequate precautions to ensure confidentiality and compliance with applicable data privacy protection laws and regulations. Appropriate technical and organizational measures to protect the personal data against unauthorized disclosures or access, accidental or unlawful destruction, or accidental loss or alteration will be put in place. Sponsor personnel whose responsibilities require access to personal data agree to keep the identity of study subjects confidential.

The informed consent obtained from the subject includes explicit consent for the processing of personal data and for the Investigator to allow direct access to his or her original medical records for study-related monitoring, audit, IRB review, and regulatory inspection. This consent also addresses the transfer of the data to other entities and to other countries. All reports and communications relating to the study subjects will identify subjects only by initials and subject identification number.

Data generated for the study will be stored by the Investigator in a limited-access file area and be accessible only to representatives of the study site, Romark, the IRB, and FDA/relevant regulatory agencies. Medical information resulting from a subject's participation in this study may be given to the subject's personal physician or to the appropriate medical personnel responsible for the subject's welfare.

#### 10.1.11. Publication and Data Sharing

Presentation and/or publication of the results of the study is encouraged provided that The Romark Institute for Medical Research is notified in advance of the author's intent and is given the opportunity to review the manuscript or abstract 45 days prior to its submission for presentation at a scientific meeting or for publication in a scientific journal. The Investigators will have complete autonomy regarding the content and wording of any abstracts, presentations, and scientific publications arising from this study, including the decision of whether or not to publish.

## 10.1.12. Key Roles and Study Governance

See Appendix 2 for a list of key personnel and contact information.

#### 11. REFERENCES

ALINIA (nitazoxanide) prescribing information. Romark, L.C., Tampa, FL, June 2019.

Allan GM, Arroll B. Prevention and treatment of the common cold: making sense of the evidence. *CMAJ* 2014 Feb 18; 186(3): 190-199.

Anderson VR, Curran MP. NTZ: A review of its use in the treatment of gastrointestinal infections. *Drugs* 2007;67:1947-67.

Arruda E, Pitkaranta A, Witek TJ, Doyle C, Hayden FG. Frequency and Natural History of Rhinovirus Infections in Adults during Autumn. *J Clin Microbio* Nov 1997; 2864-2868.

Ashton LV, Callan RL, Rao S, Landolt GA. In vitro susceptibility of canine influenza A (H3N8) virus to nitazoxanide and tizoxanide. *Vet Med Int* 2010; 2010:891010.

Backman JT, Filppula AM, Niemi M, Neuvonen PJ. Role of cytochrome P450 2C8 in drug metabolism and interactions. *Pharmacol Rev* 2016; 68:168-241.

Atkinson SK, Sadofsky LR, Morice AH. How does rhinovirus cause the common cold cough? *BMJ Open Respiratory Research* 2016;3:e000118.

Braakman I, Helenius J, Helenius A. Role of ATP and disulphide bonds during protein folding in the endoplasmic reticulum. *Nature* 1992; 356:260-62.

Braakman I, Hoover-Litty H, Wagner KR, Helenius A. Folding of influenza hemagglutinin in the endoplasmic reticulum. *J Cell Biol* 1991; 114:401-11.

Cao J, Forrest JC, Zhang X. A screen of the NIH collection small molecule library identifies potential coronavirus. *Antiviral Res* 2015; 114:1-10.

Chang CW, Li HC, Hsu CF, Chang CY, Lo SY. Increased ATP generation in the host cell is required for efficient vaccinia virus production. *J Biomed Sci* 2009; 16:80.

Doms RW, Keller DS, Helenius A, Balch WE. Role of adenosine triphosphate in regulating the assembly and transport of vesicular stomatitis virus G protein trimers. *J Cell Biol* 1987; 105:1957-69.

Fendrick AM, Monto AS, Nightengale B, Sames M. The economic burden of non-influenzarelated viral respiratory infection in the United States. *Arch Intern Med* 2003; 163(4):487-94.

Hadad GM, Abdel Salam RA, Emara S. Validated and optimized high-performance liquid chromatographic determination of tizoxanide, the main active metabolite of nitazoxanide in human urine, plasma and breast milk. *J Chromatogr Sci.* 2012;50:509-15.

Hong SK, Kim HJ, Song CS, Choi IS, Lee JB, Park SY. Nitazoxanide suppresses IL-6 production in LPS-stimulated mouse macrophages and TG-injected mice. *Int Immunopharmacol* 2012; 13:23-27.

Jacobs SE, Lamson DM, St. George K, Walsh TJ. Human Rhinoviruses. *Clin Microb Rev* 2013; 26(1):135-152.

Kirkpatrick GL. The Common Cold. *Primary Care: Clinics in Office Practice* 1996; 23(4):657-675.

Lee JH, Zhang Y, Zhao Z, Ye X, Zhang X, Wang H, Ye J. Intracellelular ATP in balance of proinflammatory and anti-inflammatory cytokines in adipose tissue with and without tissue expansion. *Int J Obes* 2017; 41:645-51.

Mirazimi A, Svensson L. ATP is required for correct folding and disulfide bond formation rotavirus VP7. *J Virol* 2000; 74:8048-52.

Piacentini S, La Frazia S, Riccio A, Pedersen JZ, Topai A, et al. Nitazoxanide inhibits paramyxovirus replication by targeting the Fusion protein folding: role of glycoprotein-specific thiol oxidoreductase ERp57. *Sci Rep* 2018; 8:10425.

Pilorge L, Chartier M, Meritet J-F, et al. Rhinoviruses as an Unprecedented Cause of Influenza-Like Illness in Pregnancy During the 2009-2010 Influenza Pandemic. *J Med Virol* 2013; 85(8):1473-7.

Powers JH, Bacci ED, Leidy NK, Poon JL, Stringer S, et al. Performance of the inFLUenza patient-reported outcome (FLU-PRO) diary in patients with influenza-like illness (ILI). *PLoS ONE* 2018 13(3):d0194180.

Rossignol JF, La Frazia S, Chiappa L, Ciucci A, Santoro MG. Thiazolides, a new class of antiinfluenza molecules targeting viral hemagglutinin at the post-translational level. *J Biol Chem* 2009; 284:29798-808.

Rossignol JF, van Baalen C. Broad-spectrum antiviral nitazoxanide inhibits ATP-dependent replication of respiratory viruses and proinflammatory cytokines [Abstract]. Presented at the 2nd International Meeting on Respiratory Pathogens. Singapore, March 7-9, 2018.

Rossignol JF. Nitazoxanide, a new drug candidate for the treatment of Middle East respiratory syndrome coronavirus. *J Infect Public Health* 2016; 9:227-30.

Rossignol JF. Nitazoxanide: A first-in-class broad-spectrum antiviral agent. *Antiviral Res* 2014; 110:94-103.

Sag D, Carling D, Stout RD, Suttles J. AMP-activated protein kinase promotes macrophage polarization to an anti-inflammatory functional phenotype. *J Immunol* 2008; 181:8633-41.

Sleeman K, Mishin VP, Guo Z, Garten RJ, Balish A, et al. Antiviral susceptibility of variant influenza A(H3N2)v viruses isolated in the United States from 2011 to 2013. *Antimicrob Agents Chemother* 2014; 58:2045-51.

St. Jude Children's Research Hospital. Infections in Immunocompromised Patients. Accessed 22 Jun 2020. Available at: https://www.stjude.org/treatment/patient-resources/caregiver-resources/infection-tips/infections-immunocompromised-patients.html

The Pirbright Institute, UK. (2018). Enterovirus. Retrieved from: http://www.picornaviridae.com/enterovirus/ enterovirus.htm

Tilmanis D, van Baalen C, Oh DY, Rossignol J-F, Hurt AC. The susceptibility of circulating human influenza viruses to tizoxanide, the active metabolite of nitazoxanide. *Antivir Res* 2017; 147:142-48.

Turner RB. Epidemiology, Pathogenesis, and Treatment of the Common Cold. *Annals of Allergy, Asthma & Immunology* 1997; 78(6):531-540.

United States Department of Labor – Bureau of Labor Statistics. CPI Inflation Calculator. Available at: https://www.bls.gov/data/inflation\_calculator.htm

van der Vries E, Stittelaar KJ, van Amerongen G, et al. Prolonged influenza virus shedding and emergence of antiviral resistance in immunocompromised patients and ferrets. *PLoS Pathog*. 2013;9(5):e1003343.

Wang M, Cao R, Zhang L, Yang X, Liu J, et al. Remdesivir and chloroquine effectively inhibit the recently emerged novel coronavirus (2019-nCoV) in vitro. *Cell Res* 2020; 30:269-71.

Wang W, Yang X, de Silanes IL, Carling D, Gorospe M. Increased AMP:ATP Ratio and AMP-activated protein kinase activity during cellular senescence linked to reduced HuR function. *J Biol Chem* 2003; 278:27016-23.

Worrall G. Common cold. Can Fam Physician 2011; 57(11):1289-1290.

Yu J, Powers JH, Vallo D, Falloon J. Evaluation of efficacy endpoints for a phase IIb study of a respiratory syncytial virus vaccine in older adults using patient-reported outcomes with laboratory confirmation. *Value Health* 2020; 23:227-35.

## APPENDIX 1. PROTOCOL REVISION HISTORY

Table 7: Protocol Revision History

| Summary of Changes | |
|---|---|
| Initial Protocol | |
| Purpose: | New protocol |
| Effective date: | July 16, 2020 |
| Amendment 1 | |
| Purpose: | <ul> <li>To revise patient selection criteria and study procedures</li> <li>To update Study Contact Information</li> <li>To correct typographical errors</li> </ul> |
| Effective Date: | December 23, 2020 |
| Change 1: | Section 1.1 Synopsis, Section 4.1 Study Design Overview Updated anticipated enrollment end from October 2020 to May 2021 |
| Change 2: | <ul> <li>Section 1.1 Synopsis, Section 5 Study Population</li> <li>Updated patient selection criteria to:</li> <li>Update inclusion criterion #3 to allow enrollment of subjects up to 72 hours from symptom onset (from 48 hours)</li> <li>Remove exclusion of subjects with oral temperature ≥100.4°F (exclusion #1)</li> <li>Added exclusion #3d, "Subjects using steroids as maintenance therapy for chronic conditions"</li> <li>Added exclusion criteria 14, "Subjects taking medications considered to be major CYP2C8 substrates. Refer to Table 6 in Section 6.5." and updated Section 6.5 Concomitant Therapy accordingly.</li> <li>Added exclusion criteria 15, "Persons with any clinical sign or symptoms suggestive of severe systemic illness with COVID-19, including the following: (a) shortness of breath at rest, (b) resting pulse ≥125 beats per minute, (c) resting respiratory rate ≥30 breaths per minute, or (d) SpO2 ≤ 93% on room air at sea level." (see also: Section 4.2.3.1 Choice of Signs and Symptoms Required for Inclusion)</li> </ul> |

| Summary of Cha | nges | |
|---|---|---|
| | Added exclusion criteri<br>infection within the pre | a 16, "Subjects known to have a diagnostic test positive for SARS-CoV-2 or influenza ceding three weeks." |
| Change 3: | Domain/Sub-domain Structure Updated study procedures to Day 6 and 7 telephone of Day 28 (±3 days) telephone Baseline and Day 22 co Subjects will complete Subjects will record ora | <ul> <li>Day 28 (±3 days) telephone contact for end-of-study safety follow-up</li> <li>Baseline and Day 22 collection of blood samples for serology testing</li> <li>Subjects will complete practice diary in the clinic at the Baseline visit</li> <li>Subjects will record oral temperature twice daily in the subject diary</li> </ul> |
| Change 4: | Specified that data for subjection criteria and proced | Section 1.1 Synopsis, Section 4.1 Study Design Overview Specified that data for subjects enrolled in concurrent study RM08-3008 (COVID-19 treatment study with the same selection criteria and procedures) with laboratory confirmed EV/RV infection at baseline will be allocated to this study for analysis and will count toward the 350 to 400 required subjects. |
| Change 5: | Section 4.1 Study Design Over Updated the randomization is Severity of Illness: Underlying Asthma, COPD Diabetes: Smoking History: | <ul> <li>tratification from:</li> <li>≤1 respiratory domain* with score ≥2 at baseline</li> <li>2 respiratory domain* with scores ≥2 at baseline</li> <li>≥3 respiratory domains* with scores ≥2 at baseline</li> <li>*For this purpose, respiratory domains shall include the following 5 FLU-PRO domains/subdomains: chest, cough, nose, throat and head.</li> </ul> |

47

| Summary of Ch | anges | |
|---|---|---|
| | Severity of Illness: | • Mild illness defined as baseline assessments of (1) at least one respiratory domain* with a baseline score ≥2 and (2) resting pulse <90 beats per minute and (3) resting respiratory rate <20 breaths per minute. |
| | | <ul> <li>Moderate illness defined as baseline assessments of (1) at least one<br/>respiratory domain* with a baseline score ≥2 and either (2) resting pulse<br/>≥90 beats per minute or (3) resting respiratory rate ≥20 breaths per minute.</li> </ul> |
| | | * For this purpose, respiratory domains shall include the following 5 FLU-PRO domains/subdomains: chest, cough, nose, throat and head. |
| | Time from onset of symptoms to | |
| | randomization: | <36 hours/≥36hours |
| | Risk of severe illness (per CDC): | <ul> <li>At Increased Risk: Subjects with COPD, Type 2 diabetes mellitus, obesity (BMI ≥30), chronic kidney disease, sickle cell disease, serious heart conditions (such as heart failure, coronary artery disease, or cardiomyopathies), asthma (moderate or severe), cerebrovascular disease, cystic fibrosis, hypertension or high blood pressure, immunocompromised state (due to immune deficiencies, HIV, use of corticosteroids, or use of other immune-weakening medications), neurologic conditions (e.g., dementia), liver disease, pulmonary fibrosis, past or present history of smoking, thalassemia, or type 1 diabetes mellitus. Subjects who are ≥65 years of age.</li> <li>Not At Increased Risk: Subjects with none of the above conditions</li> </ul> |
| Change 6: | | g the COVID-19 pandemic and is likely to enroll significant numbers of subjects |
| | | with COVID-19. Prior to database lock and unblinding, a pooled analysis of the blinded subject data will be completed to count the number of subjects with laboratory-confirmed SARS-CoV-2 infection. |
| | In the event that ≥350 subjects with that this will provide ≥90% power survival distributions between the for the Gehan rank test using SAS RM08-3005 assuming equal allocations confirmed SARS-CoV-2 will be and | h laboratory-confirmed SARS-CoV-2 infection have been enrolled, it is expected to detect a statistically significant difference in the Time to Sustained Response NTZ and placebo treatment groups [two-sided alpha=0.05, calculations performed PROC POWER (SAS 9.4) based upon data from Romark trials RM08-3004 and attion of subjects across treatment arms]. In this case, subjects with laboratory-alyzed under a separate Statistical Analysis Plan that will be signed and placed on tistical Analysis Plan will specify Time to Sustained Response (as described above) |

| Summary of Changes | |
|---|---|
| | as the primary efficacy endpoint to be analyzed at the 0.05 level and a comparison of proportions experiencing progression to severe COVID-19 illness (defined as shortness of breath at rest and SpO2≤93% on room air) using a Cochran-Maentel-Haenszel (CMH) test stratified by the randomization strata as the key secondary analysis. Day 4 and Day 10 nasopharyngeal swabs will be analyzed for the presence of SARS-CoV-2 for all subjects positive for SARS-CoV-2 at Baseline and Day 22 nasopharyngeal swabs will be analyzed if the Day 10 sample is positive for SARS-CoV-2 [analysis using Aptima® SARS-CoV-2 Assay (Hologic, Inc, San Diego, CA) as described in Section 8.2.2.2]. Proportions of subjects positive for SARS-CoV-2 at Day 4 and Day 10 will be compared across treatment groups using a CMH test stratified by the randomization strata as an exploratory analysis. Serology samples will be analyzed for quantitative IgG and IgM antibodies and descriptive statistics of the results will be presented by treatment group. Safety and pharmacokinetics will be analyzed as described in sections 9.4.2 and 9.4.3 below. |
| Change 7: | Appendix 2 Contact Information Updated contact information for Sponsor Project Management and Central Laboratory |

## APPENDIX 2. CONTACT INFORMATION

**Table 8:** Study Contact Information

| | Medical Monitors | |
|---|---|---|
| Name: | Tyledical tylomics | |
| Title: | Medical Monitor | |
| Tel.: | | |
| Fax: | | |
| E-mail: | | |
| | Sponsor Medical Affair | S |
| Name: | | |
| Title: | VP, Medical Affairs (Romark) | |
| Tel.: | | |
| Mobile: | | |
| Fax: | | |
| E-mail: | | |
| | Sponsor Project Managem | ient |
| Name: | | |
| Title: | Clinical Operations Lead | |
| Tel.: | | |
| Mobile: | | |
| Fax: | | |
| E-mail: | | |
| | Central Laboratory ( | ) |
| Name: | | |
| Title: | Project Manager | Project Manager |
| Tel.: | | |
| Fax: | | |
| E-mail: | | |
| Investigational Product Supplier | | |
| Name: | | |
| Title: | VP, Medical Affairs (Romark) | |
| Tel.: | | |
| Mobile: | | |
| Fax: | | |
| E-mail: | | |

# APPENDIX 3. LIST OF ESSENTIAL DOCUMENTS FOR THE SITE

**Table 9: List of Essential Documents** 

| 1. Investigator's Brochure and Updates 2. Signed protocol (all verisons) and amendments, if any, and sample CRF 3. Information given to subjects: • Informed consent form (all versions) • Advertisement for subject recruitment (if used) • Any other written information 4. Financial agreement between the Investigator/institution and the study Sponsor 5. Signed agreement between involved parties: • Financial disclosure of Investigator/institution and Sponsor • Confidential Disclosure Agreement of Investigator/institution and Sponsor 6. Dated, documented approval/favorable opinion of IRB on the following: • Protocol and amendments • EDC system (if applicable • Informed consent form and any revisions • Any other written information to be provided to the subjects • Advertisement for subject recruitment (if used) • Subject compensation (if any) | | Submitted | Required for<br>Study | Required<br>for Study |
|---|---|---|---|---|
| 2. Signed protocol (all verisons) and amendments, if any, and sample CRF 3. Information given to subjects: • Informed consent form (all versions) • Advertisement for subject recruitment (if used) • Any other written information 4. Financial agreement between the Investigator/institution and the study Sponsor 5. Signed agreement between involved parties: • Financial disclosure of Investigator/institution and Sponsor • Confidential Disclosure Agreement of Investigator/institution and Sponsor 6. Dated, documented approval/favorable opinion of IRB on the following: • Protocol and amendments • EDC system (if applicable • Informed consent form and any revisions • Any other written information to be provided to the subjects • Advertisement for subject recruitment (if used) • Subject compensation (if any) | Document | to IRB | Initiation | Completion |
| sample CRF 3. Information given to subjects: • Informed consent form (all versions) • Advertisement for subject recruitment (if used) • Any other written information 4. Financial agreement between the Investigator/institution and the study Sponsor 5. Signed agreement between involved parties: • Financial disclosure of Investigator/institution and Sponsor • Confidential Disclosure Agreement of Investigator/institution and Sponsor 6. Dated, documented approval/favorable opinion of IRB on the following: • Protocol and amendments • EDC system (if applicable • Informed consent form and any revisions • Any other written information to be provided to the subjects • Advertisement for subject recruitment (if used) • Subject compensation (if any) | | | | |
| Informed consent form (all versions) Advertisement for subject recruitment (if used) Any other written information Investigator/institution and the study Sponsor Signed agreement between involved parties: Financial disclosure of Investigator/institution and Sponsor Confidential Disclosure Agreement of Investigator/institution and Sponsor Confidential Disclosure Agreement of Investigator/institution and Sponsor Dated, documented approval/favorable opinion of IRB on the following: Protocol and amendments EDC system (if applicable Informed consent form and any revisions Any other written information to be provided to the subjects Advertisement for subject recruitment (if used) Subject compensation (if any) | | | | |
| Advertisement for subject recruitment (if used) Any other written information 4. Financial agreement between the Investigator/institution and the study Sponsor 5. Signed agreement between involved parties: Financial disclosure of Investigator/institution and Sponsor Confidential Disclosure Agreement of Investigator/institution and Sponsor 6. Dated, documented approval/favorable opinion of IRB on the following: Protocol and amendments EDC system (if applicable Informed consent form and any revisions Any other written information to be provided to the subjects Advertisement for subject recruitment (if used) Subject compensation (if any) | | X | | |
| Any other written information 4. Financial agreement between the Investigator/institution and the study Sponsor 5. Signed agreement between involved parties: Financial disclosure of Investigator/institution and Sponsor Confidential Disclosure Agreement of Investigator/institution and Sponsor 6. Dated, documented approval/favorable opinion of IRB on the following: Protocol and amendments EDC system (if applicable Informed consent form and any revisions Any other written information to be provided to the subjects Advertisement for subject recruitment (if used) Subject compensation (if any) | | | | |
| 4. Financial agreement between the Investigator/institution and the study Sponsor 5. Signed agreement between involved parties: • Financial disclosure of Investigator/institution and Sponsor • Confidential Disclosure Agreement of Investigator/institution and Sponsor 6. Dated, documented approval/favorable opinion of IRB on the following: • Protocol and amendments • EDC system (if applicable • Informed consent form and any revisions • Any other written information to be provided to the subjects • Advertisement for subject recruitment (if used) • Subject compensation (if any) | | | | |
| the study Sponsor 5. Signed agreement between involved parties: • Financial disclosure of Investigator/institution and Sponsor • Confidential Disclosure Agreement of Investigator/institution and Sponsor 6. Dated, documented approval/favorable opinion of IRB on the following: • Protocol and amendments • EDC system (if applicable • Informed consent form and any revisions • Any other written information to be provided to the subjects • Advertisement for subject recruitment (if used) • Subject compensation (if any) | Any other written information | | | |
| Financial disclosure of Investigator/institution and Sponsor Confidential Disclosure Agreement of Investigator/institution and Sponsor Dated, documented approval/favorable opinion of IRB on the following: Protocol and amendments EDC system (if applicable Informed consent form and any revisions Any other written information to be provided to the subjects Advertisement for subject recruitment (if used) Subject compensation (if any) | | | | |
| Sponsor Confidential Disclosure Agreement of Investigator/institution and Sponsor Dated, documented approval/favorable opinion of IRB on the following: Protocol and amendments EDC system (if applicable Informed consent form and any revisions Any other written information to be provided to the subjects Advertisement for subject recruitment (if used) Subject compensation (if any) | <ol><li>Signed agreement between involved parties:</li></ol> | | | |
| Investigator/institution and Sponsor 6. Dated, documented approval/favorable opinion of IRB on the following: • Protocol and amendments • EDC system (if applicable • Informed consent form and any revisions • Any other written information to be provided to the subjects • Advertisement for subject recruitment (if used) • Subject compensation (if any) | | | | |
| 6. Dated, documented approval/favorable opinion of IRB on the following: • Protocol and amendments • EDC system (if applicable • Informed consent form and any revisions • Any other written information to be provided to the subjects • Advertisement for subject recruitment (if used) • Subject compensation (if any) | Confidential Disclosure Agreement of | | | |
| following: Protocol and amendments EDC system (if applicable Informed consent form and any revisions Any other written information to be provided to the subjects Advertisement for subject recruitment (if used) Subject compensation (if any) | Investigator/institution and Sponsor | | | |
| <ul> <li>EDC system (if applicable</li> <li>Informed consent form and any revisions</li> <li>Any other written information to be provided to the subjects</li> <li>Advertisement for subject recruitment (if used)</li> <li>Subject compensation (if any)</li> </ul> | | | X | |
| Informed consent form and any revisions Any other written information to be provided to the subjects Advertisement for subject recruitment (if used) Subject compensation (if any) | Protocol and amendments | | | |
| Any other written information to be provided to the subjects Advertisement for subject recruitment (if used) Subject compensation (if any) | EDC system (if applicable | | | |
| subjects Advertisement for subject recruitment (if used) Subject compensation (if any) | <ul> <li>Informed consent form and any revisions</li> </ul> | | | |
| Advertisement for subject recruitment (if used) Subject compensation (if any) | | | | |
| Subject compensation (if any) | _ | | | |
| Any other documents given approval | <ul> <li>Any other documents given approval</li> </ul> | | | |
| Continuing review of the trial | Continuing review of the trial | | | |
| 7. Institutional Review Board Composition | 7. Institutional Review Board Composition | | | |
| 8. Regulatory notice of Principal Investigator and sub-<br>Investigator, FDA Form 1572 | | | | |
| Curriculum vitae and/or other relevant documents evidencing X X qualifications of Investigator and sub-Investigators | | X | X | |
| 10. Normal values/ranges and updates for medical/laboratory/ technical procedures and/or tests included in the protocol | <ol> <li>Normal values/ranges and updates for medical/laboratory/<br/>technical procedures and/or tests included in the protocol</li> </ol> | | | |
| 11. Medical/laboratory/technical procedures/tests and updates: | | | | |
| certification or | | | | |
| accreditation or | accreditation or | | | |
| established quality control and/or external quality | <ul> <li>established quality control and/or external quality</li> </ul> | | | |
| assessment or | | | | |
| other validations (where required) | other validations (where required) | | | |
| 12. Shipping records for investigational product(s) and trial-<br>related materials | | | | |
| 13. Site initiation monitoring report | 13. Site initiation monitoring report | | | |

| Document | Submitted<br>to IRB | Required for<br>Study<br>Initiation | Required<br>for Study<br>Completion |
|---|---|---|---|
| 14. Relevant communications other than site visits: | | | |
| Letters/emails | | | |
| Meeting notes | | | |
| Notes of telephone calls | | | |
| 15. Signed informed consent forms | | | X |
| 16. Source documents | | | X |
| 17. Signed, dated and completed EDC forms including documentation of EDC form corrections | | | X |
| 18. Notification by originating Investigator to Sponsor of serious adverse events and related reports | | | X |
| Notification by Investigator, where applicable, to IRB of unexpected serious adverse drug reactions and other safety information | X | | |
| 20. Notification by Sponsor to Investigator of safety information | | | |
| 21. Interim or annual reports to IRB | X | | |
| 22. Subject Screening log | | | |
| 23. Subject identification code list | | | |
| 24. Subject enrollment log | | | |
| 25. Investigational product accountability records (receipt, storage, dispensing, shipment) | | | X |
| 26. Signature sheet | | | |
| 27. Record of retained body fluids/tissue samples (if any) | | | |
| 28. Final report by Investigator/institution to IRB | X | | |

## APPENDIX 4. TOXICITY GRADING TABLES

[Derived and adapted from "Guidance for Industry: Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials", US Dept. of HHS, FDA, CDER, September 2007]

Table 10: Table for Clinical Abnormalities: Vital Signs

| Vital Signs* | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Potentially Life Threatening (Grade 4) |
|---|---|---|---|---|
| Fever (°C)** (°F)** | 38.0 – 38.4<br>100.4 – 101.1 | 38.5 – 38.9<br>101.2 – 102.0 | 39.0 – 40<br>102.1 – 104 | > 40<br>> 104 |
| Tachycardia – beats per minute | 101 – 115 | 116 – 130 | > 130 | ER visit or hospitalization for arrhythmia |
| Bradycardia – beats per minute*** | 50 – 54 | 45 – 49 | < 45 | ER visit or hospitalization for arrhythmia |
| Hypertension (systolic) – mm Hg | 141 – 150 | 151 – 155 | > 155 | ER visit or hospitalization for malignant hypertension |
| Hypertension (diastolic) – mm Hg | 91 – 95 | 96 – 100 | > 100 | ER visit or hospitalization for malignant hypertension |
| Hypotension (systolic) – mm Hg | 85 – 89 | 80 – 84 | < 80 | ER visit or hospitalization for hypotensive shock |
| Respiratory Rate – breaths per minute | 17 – 20 | 21 – 25 | > 25 | Intubation |

Subject should be at rest for all vital sign measurements.

<sup>\*\*</sup> Oral temperature; no recent hot or cold beverages or smoking.

<sup>\*\*\*</sup> When resting heart rate is between 60 – 100 beats per minute. Use clinical judgment when characterizing bradycardia among some healthy subject populations, for example, conditioned athletes.

Table 11: Table for Clinical Abnormalities: Systemic (General)

| Systemic<br>(General) | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Potentially Life Threatening<br>(Grade 4) |
|---|---|---|---|---|
| Nausea/<br>vomiting | No interference with activity or 1-2 episodes/24 hours | Some interference with activity or > 2 episodes/24 hours | Prevents daily activity,<br>requires outpatient IV<br>hydration | ER visit or hospitalization for hypotensive shock |
| Diarrhea | 2-3 loose stools or <400 gms/24 hours | 4-5 stools or 400-800 gms/24 hours | 6 or more watery stools or<br>>800 gms/24 hours or<br>requires outpatient IV<br>hydration | ER visit or hospitalization |
| Headache | No interference with activity | Repeated use of non-narcotic pain reliever >24 hours or some interference with activity | Significant; any use of narcotic pain reliever or prevents daily activity | ER visit or hospitalization |
| Fatigue | No interference with activity | Some interference with activity | Significant; prevents daily activity | ER visit or hospitalization |
| Myalgia | No interference with activity | Some interference with activity | Significant; prevents daily activity | ER visit or hospitalization |

Table 12: Table for Clinical Abnormalities: Systemic Illness

| Systemic Illness | Mild | Moderate | Severe | Potentially Life |
|---|---|---|---|---|
| | (Grade 1) | (Grade 2) | (Grade 3) | Threatening (Grade 4) |
| Illness or clinical adverse event<br>(as defined according to<br>applicable regulations) | No interference with activity | Some interference with activity not requiring medical intervention | Prevents daily activity<br>and requires medical<br>intervention | ER visit or<br>hospitalization |

The laboratory values provided in the tables below serve as guidelines and are dependent upon institutional normal parameters.

Table 13: Table for Laboratory Abnormalities: Serum

| Serum* | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Potentially Life<br>Threatening (Grade<br>4)** |
|---|---|---|---|---|
| Sodium – Hyponatremia mEq/L | 132 – 134 | 130 – 131 | 125 – 129 | < 125 |
| Sodium – Hypernatremia mEq/L | 144 – 145 | 146 – 147 | 148 – 150 | > 150 |
| Potassium – Hyperkalemia mEq/L | 5.1 – 5.2 | 5.3 – 5.4 | 5.5 – 5.6 | > 5.6 |
| Potassium – Hypokalemia mEq/L | 3.5 – 3.6 | 3.3 – 3.4 | 3.1 – 3.2 | < 3.1 |
| Chloride –mEq/L** | Asymptomatic or mild<br>symptoms; clinical or<br>diagnostic observations<br>only; intervention not<br>indicated | Moderate; minimal,<br>local or noninvasive<br>intervention indicated;<br>limiting age-appropriate<br>instrumental ADL | Severe or medically significant but not immediately life threatening; hospitalization or prolongation of existing hospitalization indicated; disabling; limiting self-care ADL | Life-threatening consequences; urgent intervention indicated |
| Glucose – Hypoglycemia mg/dL | 65 – 69 | 55 – 64 | 45 – 54 | < 45 |
| Glucose –Hyperglycemia<br>Fasting – mg/dL<br>Random – mg/dL | 100 – 110<br>110 – 125 | 111 – 125<br>126 – 200 | >125<br>>200 | Insulin requirements or hyperosmolar coma |
| Blood Urea Nitrogen<br>BUN mg/dL | 23 – 26 | 27 – 31 | > 31 | Requires dialysis |
| Creatinine – mg/dL | 1.5 – 1.7 | 1.8 – 2.0 | 2.1 – 2.5 | > 2.5 or requires dialysis |
| Calcium – hypocalcemia mg/dL | 8.0 – 8.4 | 7.5 – 7.9 | 7.0 – 7.4 | < 7.0 |
| Calcium – hypercalcemia mg/dL | 10.5 – 11.0 | 11.1 – 11.5 | 11.6 – 12.0 | > 12.0 |

Table 13: Table for Laboratory Abnormalities: Serum (Continued)

| Serum* | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Potentially Life<br>Threatening (Grade<br>4)** |
|---|---|---|---|---|
| Magnesium – hypomagnesemia<br>mg/dL | 1.3 – 1.5 | 1.1 – 1.2 | 0.9 – 1.0 | < 0.9 |
| Phosphorous – hypophosphatemia mg/dL | 2.3 – 2.5 | 2.0 – 2.2 | 1.6 – 1.9 | < 1.6 |
| CPK – mg/dL | 1.25 – 1.5 x ULN | 1.6 – 3.0 x ULN | 3.1 –10 x ULN | > 10 x ULN |
| Albumin – Hypoalbuminemia g/dL | 2.8 – 3.1 | 2.5 – 2.7 | < 2.5 | |
| Total Protein – Hypoproteinemia<br>g/dL | 5.5 – 6.0 | 5.0 – 5.4 | < 5.0 | |
| Alkaline phosphate – increase by factor | 1.1 – 2.0 x ULN | 2.1 – 3.0 x ULN | 3.1 – 10 x ULN | > 10 x ULN |
| Liver Function Tests – ALT, AST increase by factor | 1.1 – 2.5 x ULN | 2.6 – 5.0 x ULN | 5.1 – 10 x ULN | > 10 x ULN |
| Liver Function Tests – GGT** increase by factor | >ULN – 2.5 x ULN | >2.5 – 5.0 x ULN | >5.0 – 20.0 x ULN | >20.0 x ULN |
| Bilirubin – when accompanied by<br>any increase in Liver Function Test<br>increase by factor | 1.1 – 1.25 x ULN | 1.26 – 1.5 x ULN | 1.51 – 1.75 x ULN | > 1.75 x ULN |
| Bilirubin – when Liver Function<br>Test is normal; increase by factor | 1.1 – 1.5 x ULN | 1.6 – 2.0 x ULN | 2.0 – 3.0 x ULN | > 3.0 x ULN |
| Cholesterol** | ULN – 300 mg/dL | >300 – 400 mg/dL | >400 – 500 mg/dL | >500 mg/dL |
| Triglycerides – mg/dL** | 150 mg/dL – 300 mg/dL | >300 mg/dL - 500<br>mg/dL | >500 mg/dL - 1000<br>mg/dL | >1000 mg/dL |

Table 13: Table for Laboratory Abnormalities: Serum (Continued)

| Serum* | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Potentially Life<br>Threatening (Grade<br>4)** |
|---|---|---|---|---|
| HDL – mg/dL** | Asymptomatic or mild<br>symptoms; clinical or<br>diagnostic observations<br>only; intervention not<br>indicated | Moderate; minimal,<br>local or noninvasive<br>intervention indicated;<br>limiting age-appropriate<br>instrumental ADL | Severe or medically<br>significant but not<br>immediately life<br>threatening;<br>hospitalization or<br>prolongation of existing<br>hospitalization<br>indicated; disabling;<br>limiting self care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated |
| LDL – mg/dL** | Asymptomatic or mild<br>symptoms; clinical or<br>diagnostic observations<br>only; intervention not<br>indicated | Moderate; minimal,<br>local or noninvasive<br>intervention indicated;<br>limiting age-appropriate<br>instrumental ADL | Severe or medically significant but not immediately life threatening; hospitalization or prolongation of existing hospitalization indicated; disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated |

<sup>\*</sup> The laboratory values provided in the tables serve as guidelines and are dependent upon institutional normal parameters. Institutional normal reference ranges should be provided to demonstrate that they are appropriate.

Note: "ULN" is the upper limit of the normal range.

<sup>\*\*</sup> Derived from the National Institutes of Health, National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0. ADL- Activities of Daily Living refer to preparing meals, shopping for groceries or clothes, using the telephone, managing money, etc. selfcare ADL refer to bathing, dressing and undressing, feeding self, using the toilet, taking medications, and not bedridden.

Table 14: Table for Laboratory Abnormalities: Hematology

| Hematology* | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Potentially Life<br>Threatening (Grade 4) |
|---|---|---|---|---|
| Hemoglobin (Female) – gm/dL | 11.0 – 12.0 | 9.5 – 10.9 | 8.0 – 9.4 | < 8.0 |
| Hemoglobin (Female) change from<br>baseline value – gm/dL | Any decrease – 1.5 | 1.6 – 2.0 | 2.1 – 5.0 | > 5.0 |
| Hemoglobin (Male) – gm/dL | 12.5 – 13.5 | 10.5 – 12.4 | 8.5 – 10.4 | < 8.5 |
| Hemoglobin (Male) change from<br>baseline value – gm/dL | Any decrease – 1.5 | 1.6 – 2.0 | 2.1 – 5.0 | > 5.0 |
| Hematocrit - %** | Asymptomatic or mild<br>symptoms; clinical or<br>diagnostic observations<br>only; intervention not<br>indicated | Moderate; minimal,<br>local or noninvasive<br>intervention indicated;<br>limiting age-appropriate<br>instrumental ADL | Severe or medically significant but not immediately life threatening; hospitalization or prolongation of existing hospitalization indicated; disabling; limiting self-care ADL | Life-threatening<br>consequences; urgent<br>intervention indicated |
| WBC Increase - cell/mm <sup>3</sup> | 10,800 - 15,000 | 15,001 - 20,000 | 20,001 – 25, 000 | > 25,000 |
| WBC Decrease - cell/mm <sup>3</sup> | 2,500 – 3,500 | 1,500 – 2,499 | 1,000 – 1,499 | < 1,000 |
| Lymphocytes Decrease - cell/mm <sup>3</sup> | 750 – 1,000 | 500 – 749 | 250 – 499 | < 250 |
| Neutrophils Decrease - cell/mm <sup>3</sup> | 1,500 - 2,000 | 1,000 – 1,499 | 500 – 999 | < 500 |
| Eosinophils - cell/mm <sup>3</sup> | 650 – 1500 | 1501 - 5000 | > 5000 | Hypereosinophilic |
| Platelets Decreased - cell/mm <sup>3</sup> | 125,000 - 140,000 | 100,000 - 124,000 | 25,000 – 99,000 | < 25,000 |
| PT – increase by factor (prothrombin time) | 1.0 – 1.10 x ULN | 1.11 – 1.20 x ULN | 1.21 – 1.25 x ULN | > 1.25 ULN |
| PTT – increase by factor (partial thromboplastin time) | 1.0 – 1.2 x ULN | 1.21 – 1.4 x ULN | 1.41 – 1.5 x ULN | > 1.5 x ULN |

Table 14: Table for Laboratory Abnormalities: Hematology (Continued)

| Hematology* | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Potentially Life<br>Threatening (Grade 4) |
|---|---|---|---|---|
| Fibrinogen increase - mg/dL | 400 – 500 | 501 – 600 | > 600 | |
| Fibrinogen decrease - mg/dL | 150 – 200 | 125 – 149 | 100 – 124 | < 100 or associated with<br>gross bleeding or<br>disseminated<br>intravascular<br>coagulation (DIC) |

<sup>\*</sup> The laboratory values provided in the tables serve as guidelines and are dependent upon institutional normal parameters. Institutional normal reference ranges should be provided to demonstrate that they are appropriate.

Note: "ULN" is the upper limit of the normal range.

Table 15: Table for Laboratory Abnormalities: Urine

| Urine* | Mild<br>(Grade 1) | Moderate<br>(Grade 2) | Severe<br>(Grade 3) | Potentially Life<br>Threatening (Grade 4) |
|---|---|---|---|---|
| Protein | Trace | 1+ | 2+ | Hospitalization or dialysis |
| Glucose | Trace | 1+ | 2+ | Hospitalization for hyperglycemia |
| Blood (microscopic) – red blood<br>cells per high power field (rbc/hpf) | 1 – 10 | 11 – 50 | > 50 and/or gross blood | Hospitalization or<br>packed red blood cells<br>(PRBC) transfusion |

<sup>\*</sup> The laboratory values provided in the tables serve as guidelines and are dependent upon institutional normal parameters. Institutional normal reference ranges should be provided to demonstrate that they are appropriate.

<sup>\*\*</sup> Derived from the National Institutes of Health, National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0. ADL- Activities of Daily Living refer to preparing meals, shopping for groceries or clothes, using the telephone, managing money, etc. selfcare ADL refer to bathing, dressing and undressing, feeding self, using the toilet, taking medications, and not bedridden.

## APPENDIX 5. FLU-PRO DOMAIN/SUBDOMAIN STRUCTURE

